## NCT02896296

Study Number: INDV-6000-301

Title: An Open-Label, Depot Buprenorphine (RBP-6000) Treatment Extension Study in Subjects With Opioid Use Disorder

Statistical Analysis Plan Date: 06 October 2017

# **Statistical Analysis Plan**

| Sponsor: | Indivior Inc. |
|---|---|
| Protocol No: | INDV-6000-301 |
| Protocol Version<br>No./Date | Amendment 1 / 30-Sep-2016 |
| Title | An Open-Label, Depot Buprenorphine (RBP-6000) Treatment Extension Study in Subjects with Opioid Use Disorder |
| CRF Version No./Date | 5.0 / 17 Mar 2017 |
| SAP Version No./Date: | 1.0 / 06 Oct 2017 |

| Sponsor | |
|---------------------------------|-------------------------------------------|
| Sponsor Name: | Indivior Inc. |
| Biostatistics/ Title: | Associate Fellow |
| Medical/Title: | , Medical Monitor |
| Quartesian | |
| <b>Project Manager/Title:</b> | , Senior Statistical Programmer / Analyst |
| <b>Biostatistician / Title:</b> | , Manager in Biometrics |

#### INDV-6000-301

An Open-Label, Depot Buprenorphine (RBP-6000) Treatment Extension Study in Subjects with Opioid Use Disorder

Final Version 1.0: October 6, 2017

# Confidentiality Statement

The information contained in this document is privileged and confidential. Do not copy, circulate, or otherwise distribute without written authorization from Indivior Inc.

# **<u>TABLE OF CONTENTS</u>**

| Statistic | cal Analysis Plan | 1 |
|---|---|---|
| 1.0 | TITLE PAGE | 2 |
| 2.0 | TABLE OF CONTENTS | 1 |
| 3.0 | LIST OF ABBREVIATIONS | 2 |
| 4.0 | INTRODUCTION | 6 |
| 5.0 | OBJECTIVE | 8 |
| 6.0 | SUBJECT POPULATIONS AND TREATMENT GROUPS 6.1 Screened Population. 6.2 Safety Analysis Set | 9 |
| | 6.3 Treatment Groups | |
| 7.0 | SUBJECT DISPOSITION | 10 |
| 8.0 | PROTOCOL DEVIATIONS | 1 |
| 9.0 | DEMOGRAPHICS AND OTHER BASELINE CHARACTERISTICS 9.1 Substance use history 9.2 Medical History 9.3 Prior and Concomitant Medications | 12<br>12 |
| 10.0 | EXTENT OF EXPOSURE AND TREATMENT COMPLIANCE | 16 |
| 11.0 | Exploratory EFFICACY ANALYSES | |
| 12.0 | SAFETY ANALYSES | 20<br>21<br>22<br>22<br>22<br>22<br>22 |

| Indivior | Inc. | | Page 2 |
|---|---|---|---|
| | 10.0 | 12.1.12 Psychiatry History Topic of Special Interest | |
| | 12.2 | Clinical Laboratory Parameters | |
| | | 12.2.1 Hematology | |
| | | 12.2.3 Urinalysis | |
| | 12.3 | Vital Signs | |
| | 12.3 | Other Safety Parameters | |
| | 12.7 | 12.4.1 Suicidality | |
| | | 12.4.2 Local Injection Site Evaluation | |
| | | 12.4.3 Local Injection Site Tolerability | |
| | | 12.4.4 Injection Site Pain. | |
| | | 12.4.5 Other Safety Variables | |
| | 12.5 | Independent Drug Counseling/Behavioural Therapy | 28 |
| 13.0 | POOL E | D ANALYSES | 20 |
| 13.0 | TOOLL | D ANALIGES | 29 |
| 14.0 | SUBGR | ROUP ANALYSES | 30 |
| 15.0 | неліт | TH OUTCOME ANALYSES | 31 |
| 13.0 | TILALI | II OU ICOME ANALI SES | |
| 16.0 | PLASM | IA CONCENTRATION ANALYSES | 32 |
| 17.0 | INTERI | IM ANALYSIS | 33 |
| 18.0 | DETER | MINATION OF SAMPLE SIZE | 34 |
| 19.0 | COMPU | UTER METHODS | 35 |
| 20.0 | DATA | HANDLING CONVENTIONS | 36 |
| | 20.1 | Reference Dates and Analysis Periods | |
| | 20.2 | Analysis visits and Other Definitions | |
| | 20.3 | Derived Efficacy Variables | |
| | 20.4 | Repeated or Unscheduled Assessments of Safety Parameters | |
| | 20.5 | Missing Date of Investigational product | |
| | 20.6 | Missing Severity and relationship to Study Drug in Adverse Events | |
| | 20.7 | Missing Date Information for Adverse Events | |
| | 20.8 | Missing Date Information for Concomitant Medications | |
| | 20.9 | Character Values of Clinical Laboratory Parameters AND other Laborator | - |
| | | Imputation rules | 41 |
| | 20.10 | C-SSRS DATA IMPUTATION | 41 |
| 21.0 | CHANG | GES TO ANALYSES SPECIFIED IN PROTOCOL | 42 |
| 22.0 | REFER | ENCES | 43 |
| 23.0 | Append | iix | 44 |
| | 23.1 | Appendix 1: List of Preferred Terms from Standard MedDRA Queries for | Adverse |
| | | Events of Special Interest | 44 |
| | List of I | Preferred Terms for Psychiatric History | 44 |
| [INDV- | 6000-301 | I] SAP v 1.0 | October 6, 2017] |

| Indivior Inc. | Page 3 |
|---|---|
| Customized MedDRA Query (CMQ) List of Preferred Terms for Drug Related Hepatic | |
| Disorders | 51 |
| CMQ List of Preferred Terms for Injection Site Reaction | 54 |
| CMQ List of Preferred Terms for CNS Depression | 55 |
| CMQ List of Preferred Terms for Respiratory Depression/Respiratory Failure | 56 |
| CMQ List of Preferred Terms for Orthostatic Hypotension | 57 |
| CMQ List of Preferred Terms for Withdrawal Symptoms | 57 |
| CMQ List of Preferred Terms for Acute Pancreatitis | 58 |
| 23.2 Appendix 2: List of CYP3A4 Inhibitor Medications | 58 |
| 23.3 Appendix 3: Tables, Figures and Listings | 60 |

# 3.0 <u>LIST OF ABBREVIATIONS</u>

| AE | Adverse Event |
|---|---|
| ALP | Alkaline Phosphatase |
| ALT | Alanine Aminotransferase |
| AST | Aspartate Aminotransferase |
| ВМІ | Body Mass Index |
| CDF | Cumulative Distribution Function |
| CNS | Central nervous system |
| CRF | Case Report Form |
| CTMS | Clinical Trials Management System |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| ECG | Electrocardiogram |
| EOS | End of Study |
| ET | Early Termination |
| GGT | Gamma-glutamyl Transpeptidase |
| HDL-C | High-density lipoprotein - Cholesterol |
| IA | Interim Analysis |
| ICF | Informed Consent Form |
| IDC | Individual Drug Counseling |
| LDH | Lactate dehydrogenase Medical Dictionary for Regulatory Activities |
| MedDRA | Medical Dictionary for Regulatory Activities |
| ОТС | Over The Counter |
| PDV | Protocol Deviation |
| PT | Preferred Term |
| OUD | Opioid Use Disorder |
| SAP | Statistical Analysis Plan |
| SAE | Serious Adverse Event |
| SC | Subcutaneous |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| SDTMIG | Study Data Tabulation Model Implementation Guide |
| SI | International System |
| SOC | System Organ Class |
| SUSAR | Suspected Unexpected Serious Adverse Event |
| TBIL | Total Bilirubin |
| TEAE | Treatment-Emergent Adverse Event |
| TFLs | Tables, Listings, and Figures |
| UDS | Urine Drug Screen |

| ULN | Upper Limit of Normal |
|---------|-------------------------------------------|
| VAS | Visual Analog Scale |
| WHODRUG | World Health Organization Drug Dictionary |

#### <u>4.0</u> <u>INTRODUCTION</u>

This statistical analysis plan (SAP) describes the statistical methods to be used during the final reporting and analyses of data collected for the full study (Protocol INDV-6000-301).

This SAP should be read in conjunction with the study protocol and case report form (CRF). This version of the plan has been developed using the protocol dated 30SEP2016 and CRF dated 17Mar2017.

This is a multicenter, open-label, RBP-6000 treatment extension study in which approximately 300 subjects diagnosed with moderate to severe Opioid Use Disorder (OUD) will be enrolled. Enrollment is defined as the first dose of RBP-6000 administered for this study. Only subjects who have completed the End of Study (EOS) procedures for Study RB-US-13-0003, have signed the INDV-6000-301 informed consent form (ICF), and meet all enrollment criteria will be considered for inclusion in this study.

The Institutional Review Board (IRB) approved ICF may be shared with the potential subject up to 2 months before the EOS Visit for Study RB-US-13-0003 to discuss this study as a possible treatment option. However, the ICF for Study INDV-6000-301 must not be signed until all assessments for the RB-US-13-0003 EOS Visit are complete.

The RB-US-13-0003 EOS assessments completed at the EOS Visit will serve as part of the screening assessments for this study. In addition, medical history will be collected, height measured, and subjects will be requested to complete a Columbia Suicide Severity Rating Scale (C-SSRS) baseline survey.

On Day 1 (the date of the first injection), eligible subjects will receive a subcutaneous (SC) injection of RBP-6000. For each injection, subjects may receive either 100 mg or 300 mg of RBP-6000 (to be referred to as 100/300 Flex for the remainder of this document), based on the medical judgment of the investigator. Following RBP-6000 injection, vital signs and the injection site will be assessed. The injection site will be assessed by the site for pain, tenderness, erythema/redness, induration and swelling using a 5-point severity scale (the Injection Site Grading Scale). In addition, the subject will assess their own injection site pain using a visual analog scale (VAS) (referred to as the Injection Site Pain VAS). Before departing the site, the subject will also be assessed for adverse events (AEs) and use of concomitant medications.

Subjects will not be permitted to receive supplemental buprenorphine during the RBP-6000 treatment period (Day 1 to EOS/ET Visit). Subjects who require supplemental buprenorphine pharmacotherapy during the RBP-6000 treatment period will be withdrawn from the study and referred for appropriate treatment.

Subjects will return to the site for monthly injection visits every 28 days (-2 / +7 days) for a total of up to 6 injections. Subjects are not required to complete all 6 injections and may choose to "early terminate" (ET) the study at any time.

At each subsequent visit (Injection Visits 2 through 6) the following procedures and assessments will be performed: urine pregnancy test for all female subjects who are of childbearing potential before each injection; evaluation of previous injection site for potential reaction and evidence of attempts to remove the depot; collection of vital signs pre- and post-injection; RBP-6000 injection; urine drug screen (UDS); C-SSRS since last visit, counseling (manual-guided behavioral therapy); local injection site grading; subject self-assessment of injection site pain (Injection Site Pain VAS); use of concomitant medications; and assessment for AEs. Laboratory tests (hematology, chemistry and urinalysis) may be requested by the investigator on an ad-hoc basis as necessary to further examine any AEs.

Alternative treatment options should be assessed at least two months before EOS at each visit, however it is recommended where possible to assess at every visit.

At the EOS/ET Visit, the following procedures and assessments will be performed: urine pregnancy test for all female subjects who are of childbearing potential; evaluation of previous injection site for potential reaction and evidence of attempts to remove the depot; vital sign measurements; UDS; C-SSRS since last visit, counseling (manual-guided behavioral therapy); use of concomitant medications; assessment for AEs; brief physical exam; body weight measurement (to determine a subject's body mass index [BMI]); hip and waist circumference measurement (to determine a subject's hip-to-waist ratio); and laboratory tests (hematology, chemistry, urinalysis).

Approximately 4 weeks after EOS/ET Visit, all subjects should be contacted by telephone or face-to-face visit safety follow-up assessment of AEs and use of any concomitant medications.

## 5.0 OBJECTIVE

Indivior is developing RBP-6000, a long-acting formulation of buprenorphine for monthly subcutaneous (SC) injection, for the treatment of Opioid Use Disorder (OUD).

The objective is to provide ongoing treatment with RBP-6000 and safety monitoring for subjects who complete the RB-US-13-0003 study and for whom a new treatment venue has not been identified or arranged.

# 6.0 SUBJECT POPULATIONS AND TREATMENT GROUPS

#### 6.1 SCREENED POPULATION

The Screened Population Set includes any subject who signed the informed consent form.

#### 6.2 SAFETY ANALYSIS SET

The Safety Analysis Set consists of all subjects who received at least one dose of RBP-6000.

#### 6.3 TREATMENT GROUPS

There is only one treatment group in the trial and all subjects will be labeled with "RBP-6000 (100/300 mg Flex)".

6000-301 Page 10

#### **<u>7.0</u>** <u>SUBJECT DISPOSITION</u>

The number and percentage of subjects screened and screen failures, if any, will be summarized.

The number and percentage of subjects who entered the RBP-6000 treatment period (i.e., Treatment Period, and see definition in Section 20.1), and who completed the study will be presented, together with the number and percentage of subjects who prematurely discontinued from the RBP-6000 treatment period along with reasons for study discontinuation will be summarized.

In summary, it is that the following number and percentage of subjects will be presented:

- o All subjects who were considered screen-failures
- o All subjects who entered the RBP-6000 treatment period (i.e., Treatment Period, and see definition in Section 20.1)
  - All subjects who completed the study
  - All subjects who prematurely discontinued from the RBP-6000 treatment period along with reasons for study discontinuation.

The number and percentage of subjects included in each analysis set will be presented.

A listing of the inclusion/exclusion reasons for screen failures will be provided, if any.

## 8.0 PROTOCOL DEVIATIONS

A listing of important protocol deviations (PDV) will be presented by subject using the Safety Analysis Set. An important deviation is defined as:

- Subject was deemed eligible for the study but did not meet inclusion/exclusion criteria
- Consent was not obtained from the subject

#### 9.0 DEMOGRAPHICS AND OTHER BASELINE CHARACTERISTICS

Demographic and baseline characteristics (sex, ethnicity, race, age [years and categories of  $\geq 18$ - $<30, \geq 30$ - $<45, \geq 45$ - $<60, \geq 60$  and  $\geq 65$ ], weight [kg], height[cm], waist[cm], hip[cm], waist-to-hip ratio and body mass index [BMI; kg/m2]) will be summarized using descriptive statistics for subjects in the Safety Analysis Set. Qualitative variables (sex, ethnicity, race, age categories, BMI categories) will be summarized using frequencies while quantitative variables (age, weight, height, BMI, waist, hip and waist-to-hip ratio) will be summarized using mean, SD, median, minimum, and maximum. Demographic and baseline data will also be listed for all subjects.

#### 9.1 SUBSTANCE USE HISTORY

Substance use history will be presented by substance and previous use for subjects in the Safety Analysis Set. Tobacco use [never, former, current], caffeine use [never, former, current], alcohol use [never, former, current]) will be summarized using descriptive statistics for subjects in the Safety Analysis Set. Qualitative variables (tobacco use, caffeine use, alcohol use) will be summarized using frequencies.

#### 9.2 MEDICAL HISTORY

Medical history will be coded using Medical Dictionary for Regulatory Activities (MedDRA) version 19.0 and summarized by the number and percentage of subjects in each System Organ Class (SOC), Preferred Term (PT) and in the Safety Analysis Set. Subjects will be counted only once for each PT, only once at the System Organ Class (SOC), and only once at subject level for the counting of total number of subjects with a medical history term. Counts will be presented in descending frequency unless otherwise specified.

Listings of medical history events for each subject will be provided.

#### 9.3 PRIOR AND CONCOMITANT MEDICATIONS

Prior and concomitant medications will be categorized by preferred name and drug category class (CMCLAS, ATC level 4 class per World Health Organization Drug Dictionary [WHODRUG]); and will be summarized for the Safety Analysis Set. The number and percentage of subjects using each medication will be displayed together with the number and percentage of subjects using at least one medication.

Prior medications rolling over from prior studies will be considered for both prior and concomitant medications in this study.

#### Prior Medications

For a subject in the Safety Analysis Set, prior medications will include any medication taken within 28 days prior to subject's first dose of RBP-6000 in the INDV-6000-301 study.

Concomitant medications are defined as prescribed medications and Over The Counter (OTC) preparations, including herbal preparations and vitamins, other than RBP-6000.

All prior medications will be presented in separate listing for the Safety Analysis Set.

A summary of all concomitant medications taken from Day 1 to last dose + 28 days will be presented as during RBP-6000 dosing for the Safety Analysis Set.

A summary of all concomitant medications taken from the last dose + 29 days to the last recorded assessment will be presented as post RBP-6000 dosing for the Safety Analysis Set.

A listing of all subject's concomitant medications during RBP-6000 dosing and post RBP-6000 dosing will be listed separately.

After imputing the incomplete start/end date of non-study medications (as described in Section 20.8), the determination of concomitant medication during vs. post RBP-6000 dosing follows the rules in the Table 1 below.

Table 1: Determination of Concomitant Medication during vs. Post RBP-6000 doing

| | | Start date of Non-Study Medication | | | |
|---|---|---|---|---|---|
| | | missing | Prior to day 1 | from Day 1 to last<br>dose +28 days<br>(inclusive) | Post last<br>dose+28 days |
| End date of non-study medication | missing | During <sup>1</sup> ,<br>Post <sup>2</sup> | During, Post | During, Post | Post |
| | from Day 1 to last<br>dose +28 days<br>(inclusive) | During | During | During | Data error |
| | Post last dose+28 days | During,<br>post | During, post | During, post | post |

<sup>&</sup>lt;sup>1</sup> during RBP-6000 dosing. <sup>2</sup> post RBP-6000 dosing

#### **CNS Depressants**

If a subject satisfies any of the three criteria below, then the subject is classified as taking a CNS Depressant

# Criterion 1: [INDV-6000-301] SAP Version 1.0

RBP-6000


Subject with concomitant medication and its class (CMCLAS) in ('BENZODIAZEPINE RELATED DRUGS' 'BENZODIAZEPINE DERIVATIVES' 'DIAZEPINES, OXAZEPINES, THIAZEPINES AND OXEPINES' 'OTHER HYPNOTICS AND SEDATIVES' 'PHENOBARBITAL'). Defined in the later section (CNS Depressant Medication Categories)

#### Criterion 2:

Subject with substances 'Barbiturates' or 'Benzodiazepine' detected positive in Urine Drug Screen during the Treatment Period.

#### **CNS Depressant Medication Categories**

#### Benzodiazepine-related drugs

If the Concomitant medication class is "BENZODIAZEPINE RELATED DRUGS" or detection of substances "Benzodiazepine" positive in Urine Drug Screen positive during the Treatment Period, then it is derived as Benzodiazepine related drugs.

#### Benzodiazepine derivatives

If the Concomitant medication class contains ("BENZODIAZEPINE DERIVATIVES", "DIAZEPINES, OXAZEPINES, THIAZEPINES AND OXEPINES") during the Treatment Period then it is derived as Benzodiazepine Derivatives.

#### Other Hypnotics and Sedatives

If the Concomitant medication class is ("OTHER HYPNOTICS AND SEDATIVES") during the Treatment Period, then it is derived as Other Hypnotics and Sedatives.

#### Phenobarbital and Derivatives

If the Concomitant medication class is "PHENOBARBITAL" during RBP-600 dosing or detection of substances Barbiturates positive in Urine Drug Screen during the Treatment Period, then it is derived as Phenobarbital and Derivatives.

Summary of subjects who have taken CNS depressant medications during RBP-6000 dosing (from Day 1 to last dose + 28 days) be provided. CNS depressant medications can be indemnified from two sources in this study: Concomitant medications or Urine Drug Screen as in the table below (Table 2).

Table 2: Summary of Subjects Who Have Taken CNS Depressant Medications During RBP-6000 Dosing

Any CNS depressant (from Concomitant medications) taken with a start date after Day 1 to last dose + 28 days

Benzodiazepine-related Drugs

**Benzodiazepines Derivatives** 

Other Hypnotics and Sedatives

Phenobarbital and Derivatives

Any positive CNS depressant (from UDS) during the treatment period

**Barbiturate Positive** 

**Benzodiazepines Positive** 

Preferred terms at drug class ATC level 3 of drug categories Benzodiazepine-related Drugs, Benzodiazepines Derivatives, Other Hypnotics and Sedatives and Phenobarbital and Derivatives will be summarized in the safety analysis set (see Appendix 1 for the list of CNS depressant medications).

A separate table for CNS depressant medications will be summarized for post RBP-6000 dosing

#### **CYP3A4 Inhibitor Medication Categories**

The following four categories (Unclassified, Weak, Moderate and Strong) are used from Appendix 2 containing Generic/Brand name of the CYP3A4 Inhibitor medication and its categories.

Preferred terms at drug class ATC level 3 of CYP3A4 Inhibitor Medications (Unclassified, Weak, Moderate or Strong inhibitors) during RBP-6000 dosing and post RBP-6000 dosing will be summarized in separate tables.

#### 10.0 EXTENT OF EXPOSURE AND TREATMENT COMPLIANCE

#### 10.1 EXTENT OF EXPOSURE

Exposure duration is defined as the date of last injection + 28 days - the date of first injection +1.

A summary of the exposure to RBP-6000 during the treatment period will be summarized by visit and dosage for the Safety Analysis Set. A listing of RBP-6000 exposure (administration/dispensation) will be provided.

The duration of exposure in 4 week intervals (i.e., 0 - <4 weeks, 4 - <8 weeks through 20 - <24 weeks and >= 24 weeks), total number of RBP-6000 doses received, the total number of actual doses as a categorical summary will be presented by dose received in the Safety Analysis Set. RBP-6000 exposure data will also be listed detailing the dose of RBP-6000 received at each injection and days since last injection. Besides, the cumulative frequency distribution will be tabulated by categories of >0 weeks, >=4 weeks through >=24 weeks.

The number of subjects who had an early surgical removal of the RBP-6000 depot will be presented for the Safety Analysis Set and by dose level (i.e., either 100 mg or 300 mg). Early surgical removal of the study drug depot data including the reason and surgical removal date and time will be listed, if surgical removal of the RBP-6000 depot occurs within the study.

#### 10.2 INJECTION DOSE AND VISIT COMPLIANCE

Number and percentage of subjects with injection administrated at each visit will be tabulated in the Safety Analysis Set. Cumulative frequency distribution of injections will be summarized.

Dose level frequency distribution (either 100 mg or 300 mg) at each visit will be summarized. Dose level over time during the treatment period for subjects who received 100 mg at the first injection and 300 mg at the first injection will be summarized respectively in the Safety Analysis Set.

Dose modification and its reason (adverse event, lower dose strategy or other) over time will be summarized and its distribution per visit will be plotted using stacked-bar plot. Listing of all subjects who experienced dose adjustments should be provided, including dose prior to and after dose adjustment, and reason for dose adjustment.

Days since last injection will be summarized in the safety analysis set and the distribution of the relative study days of injections will be plotted and listed.

#### 11.0 EXPLORATORY EFFICACY ANALYSES

#### 11.1 URINE DRUG SCREEN (UDS)

The urine sample collected at Screening visit will be tested for drugs listed in the Table 3. The drugs classified as opioids are identified in the same table.

Table 3: Opioid Drug Classification in Urine Drug Screen at Screening Visit.

| Drug | Opioid? |
|--------------------------------------|---------|
| Amphetamine | No |
| Barbiturates | No |
| Benzodiazepine | No |
| Benzoylecgonine (Cocaine metabolite) | No |
| Cannabinoids | No |
| Opiates | Yes |
| Codeine | Yes |
| Hydrocodone | Yes |
| Hydromorphone | Yes |
| Methadone | Yes |
| Morphine | Yes |
| Oxycodone | Yes |
| Oxymorphone | Yes |
| Methamphetamine | No |
| Phencyclidine | No |

At Screening, specific substances were confirmed once the test for Opiates was positive. The UDS for Opioids at Screening will be defined as follows:

The UDS for Opioids is Non-negative at Screening if at least one UDS result (listed in Table ) is positive;

The UDS for Opioids is Negative at Screening, if all non-missing UDS results for opioids are negative.

If all UDS measurements for opioids are missing at Screening, the UDS for Opioids will be classified as missing; then be imputed as Non-negative; and be flagged as "Non-Responder Imputation".

The urine sample collected at visits in the Treatment Period will be tested for drugs listed in the Table 4. The drugs classified as opioids are identified in the same table.

Table 4: Opioid Drug Classification in Urine Drug Screen at visits in the Treatment Period

| Drug | Opioid? |
|--------------------------------------|---------|
| Amphetamine | No |
| Barbiturates | No |
| Benzodiazepine | No |
| Benzoylecgonine (Cocaine metabolite) | No |
| Cannabinoids | No |
| Opiates | Yes |
| Methadone | Yes |
| Oxycodone | Yes |
| Methamphetamine | No |
| Phencyclidine | No |

Different from Screening Visit, specific opiate substances were not confirmed when the Opiates test was positive. Samples were tested for Oxycodone and Methadone separately from the Opiates test.

The UDS for Opioids at visits in the Treatment Period will be defined as follows: The UDS for Opioids is Non-negative at visits in the Treatment Period if at least one UDS result (listed in Table 4; either the Opiates test, or individual test for Methadone or individual test for Oxycodone) is positive;

The UDS for Opioids is Negative at visits in the Treatment Period, if all non-missing UDS results for opioids are negative.

If all UDS measurements for opioids are missing at visits in the Treatment Period, the UDS for Opioids will be classified as missing; and then be imputed as Non-negative; and be flagged as "Non-Responder Imputation".

The percentage of UDS Negative for Opioids during the Treatment Period (i.e., only for scheduled visits in the Treatment Period) will be calculated by subject, as the number of visits with UDS Negative for Opioid for that subject divided by the number of scheduled visits during the Treatment Period. Note that this means that subject missing UDS for Opioids for any scheduled visit will be classified as Non-negative for that visit. The subject-specific percentage of UDS Negative for opioids will be summarized using Descriptive statistics (n, mean (SD), median, min and max). The cumulative distribution function (CDF) will be tabulated for the following categories: >=0%, >=10%, >=20% through 100%.

A subject is classified as 'treatment success', if his/her percentage of UDS Negative for Opioids is >=80% during the Treatment Period. The Number and percentage of treatment successes will be summarized

The number and percentage of subjects with UDS Negative for Opioids by visit at Screening/Baseline or during the Treatment Period will be summarized. The denominator /INDV-6000-301] SAP Version 1.0 October 6, 2017

RBP-6000 INDV-6000-301

Page 19

of the percentage will be the number of subjects in the Safety Analysis Set. Additionally, the percentage of subjects with UDS Negative for Opioids by visit will also be calculated using the available data approach, where the subjects missing UDS for Opioids for a visit will be excluded from the denominator of the percentage for that visit.

The number and percentage of subjects with positive UDS results will be summarized for the substances tested or for Opiates test during the Treatment Period. The subject will be classified as positive for available substance/Opiates if the UDS result for that substance/Opiates is reported as positive at least once during the Treatment Period. Note that the subjects are only counted once for each substance or for the Opiates test.

All drugs detected in the UDS tests (either Negative or Non-negative) for each subject, for all visits (scheduled or unscheduled), will be listed.

#### 12.0 SAFETY ANALYSES

All analyses will be conducted by Analysis Period (s) over time at each analysis visit or overall in the Safety Analysis Set. Please see definition for Analysis Period and Analysis Visit in Section 20.1 and 20.2 respectively.

The following variables will be evaluated to assess the safety and tolerability of RBP-6000:

- Incidence of treatment-emergent adverse events (TEAEs).
- Changes in clinical laboratory results.
- Vital sign measurements.

Other Safety Variables are:

- Medical history.
- Urine pregnancy test.
- Suicidality using the C-SSRS.
- Prior and concomitant medications.
- Local injection site tolerability (e.g., injection site grading).
- Injection site pain using a subject-reported VAS.
- Weight, BMI, waist circumference, hip circumference and waist-to-hip ratio.
- Behavioral therapy.

#### 12.1 ADVERSE EVENTS

#### 12.1.1 Adverse Events

Imputation rules for AE (for determination of TEAE only) start date are in Section 20.7.

#### **Treatment-emergent Adverse Events (TEAEs)**

TEAEs are those that started following the first dose of RBP-6000 and before the Treatment End Date (the maximum of the date of the end-of-study/ Early Termination (EOS/ET) visit and the date of last injection + 28 days) in this study, or were present prior to the first dose of RBP-6000 regardless of causality and increased in severity within the treatment period (defined in section 20.1) AEs include those events that are ongoing at the time a subject rolls-over from the RB-US-13-0003.

#### **Treatment-related Adverse Events**


A summary of TEAEs will be presented for the Safety Analysis Set, including the number and percentage of subjects reporting at least one TEAE, the number and percentage of subjects with the following:

- Related TEAEs
- SAEs
- Related SAEs
- TEAEs with an outcome of death
- TEAEs
- Severe TEAEs
- TEAEs leading to RBP-6000 discontinuation

A breakdown of the number and percentage of subjects reporting each TEAE categorized by SOC and PT coded per the MedDRA dictionary version 19.0 will be presented in the Safety Analysis Set. Note that counting will be by subject not by event and subjects will be only counted once within each SOC or PT.

A further tabulation of events experienced by  $\geq 5\%$  of subjects by SOC and PT will be presented for the Safety Analysis Set. If there are no TEAEs experienced  $\geq 5\%$  of subjects by any PT, this table will be empty.

A summary of events reported, categorized by severity, will also be provided. Subjects with multiple events within a SOC or PT will be counted under the category of their most severe event within that SOC or PT. A further tabulation of severe AE/TEAEs will be presented by SOC and PT.

Additionally, treatment-related AEs/TEAEs will be summarized by maximum severity (mild, moderate, or severe). A breakdown of severe treatment-related AEs/TEAEs by SOC and PT will be provided.

All AEs (including non-TEAEs) recorded on the CRF will be listed.

#### 12.1.2 Serious Adverse Events

SAEs and treatment-related SAEs will be summarized separately by SOC and PT for the Safety Analysis Set.

All SAEs recorded on the CRF will be listed for all subjects.

#### 12.1.3 Adverse Events Leading to Discontinuation

A summary of AEs/TEAEs and treatment-related AEs/TEAEs leading to discontinuation (defined as an event with an outcome of 'drug withdrawn' in the CRF) will be provided, grouped by SOC and PT, for the Safety Analysis Set. Supportive listings will be provided.


All AEs leading to discontinuation recorded on the CRF will be listed. Additionally, TEAEs leading to dose reduction will be listed.

#### **12.1.4** Deaths

A table presenting the number and percentage of subjects who died during the Treatment Period will be presented for the Safety Analysis Set, respectively. Deaths occurring in the study will also be listed for all screened subjects, if death occurs within the study.

#### 12.1.5 Potentially Pertaining to Drug Withdrawal Symptoms

A summary of TEAEs potentially pertaining to drug withdrawal during the Treatment Period, as defined in Appendix 1, will be summarized by SOC and PT for the Safety Analysis Set.

Additionally, A summary table of Adverse Events potentially pertaining to drug withdrawal during the Safety Follow-up Period will be used to tabulate AEs related to drug withdrawal symptoms in the Safety Follow-Up period after EOS/ET visit, if any.

#### 12.1.6 Potentially Pertaining to Injection Site Reactions

A summary of TEAEs potentially pertaining to injection site reactions, as defined in Appendix 1, will be summarized by SOC and PT for the Safety Analysis Set.

#### 12.1.7 Hepatic Disorders Topic of Special Interest

A summary of TEAEs potentially related to hepatic disorders, as defined in Appendix 1, will be summarized by SOC and PT for the Safety Analysis Set.

#### 12.1.8 Central Nervous System Depression Topic of Special Interest

A summary of TEAEs related to Central Nervous System Depression, as defined in Appendix 1, will be summarized by SOC and PT for the Safety Analysis Set.

#### 12.1.9 Respiratory Depression Topic of Special Interest

A summary of TEAEs related to respiratory depression, as defined in Appendix 1, will be summarized by SOC and PT for the Safety Analysis Set.

#### 12.1.10 Acute Pancreatitis Topic of Special Interest

A summary of TEAEs related to acute pancreatitis as defined in Appendix 1, will be summarized by SOC and PT for the Safety Analysis Set.

## 12.1.11 Orthostatic Hypotension Topic of Special Interest

A summary of TEAEs related to orthostatic hypotension, as defined in Appendix 1, will be summarized by SOC and PT for the Safety Analysis Set.

## 12.1.12 Psychiatry History Topic of Special Interest

A summary of TEAEs regarding psychiatry history, as defined in Appendix 1, will be summarized by SOC and PT for the Safety Analysis Set.

#### 12.2 CLINICAL LABORATORY PARAMETERS

Laboratory data will be reported using International System (SI) units (and using original units for some parameters if necessary) as collected by the central laboratory. Unless otherwise specified, all continuous laboratory data will be summarized using descriptive statistics (n, mean, SD, median, min and max) for each scheduled study assessment as well as change from baseline and percentage change from baseline [if applicable] by parameter class (hematology, chemistry, and urinalysis). All laboratory assessments include a baseline summary as defined in Section 20.2 unless otherwise indicated. Hematology chemistry and urinalysis data will be summarized by displaying shifts from baseline value to EOS/ET visit. All laboratory assessments will be listed by panel with the corresponding normal ranges for each parameter. Screening laboratory tests will also be listed.

The peak total bilirubin [x ULN] vs. peak aspartate aminotransferase (or peak alanine aminotransferase) [x ULN] on a log/log scale during the Treatment Period will be plotted in the Safety Analysis Set. And the box plot to access clinical liver safety data by maximum change from baseline during the Treatment Period will be plotted for lab tests ALT, AST and total bilirubin.

Summary of potential hepatotoxicity for serum chemistry by type of criterion (shown in Table 5) and by analysis visit and at any time post baseline will be tabulated for the Safety Analysis Set. For "Any time post baseline", a subject will be classified to their highest/worst applicable toxicity grade per criterion, among the post baseline visits including unscheduled visits, and be counted only once in the category corresponding to the worst grade. For subjects who met the criteria for potential hepatotoxicity (any time post baseline), their test results for ALT, AST, TBIL, ALP during study (i.e., at all scheduled and unscheduled visit) will be provided in a listing.

Table 5: Criteria for Potential Hepatotoxicity Laboratory Value

| Criteria |
|-------------------------------------------------------|
| $ALT > 3 \times ULN \text{ to } < 5 \times ULN$ |
| $ALT \ge 5 \times ULN \text{ to } < 8 \times ULN$ |
| $ALT \ge 8 \times ULN$ |
| $AST > 3 \times ULN \text{ to } < 5 \times ULN$ |
| $AST \ge 5 \times ULN \text{ to } < 8 \times ULN$ |
| $AST \ge 8 \times ULN$ |
| ALT & AST $> 3$ x ULN to $< 5$ x ULN |
| ALT & AST $\geq$ 5 x ULN to $<$ 8 x ULN |
| ALT & AST $\geq 8 \times ULN$ |
| TBIL $> 2$ x ULN to $< 5$ x ULN |
| TBIL $\geq 5 \times ULN$ |
| HYs Law: (all must be met to meet Potential Hy's law) |
| ALT or AST > 3 x ULN |
| TBIL > 2 x ULN |
| ULN < Alkaline phosphatase (ALP) < 2xULN |

#### 12.2.1 Hematology

Parameters include hematocrit, hemoglobin, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, mean corpuscular volume, platelet count (available at EOS/ET only), red blood cell count and white blood cell count with differential. Visits include Screening (or EOS Visit RB-US-13-0003) and Day 169 Week 25 (EOS INDV-6000-301) /ET visit.

#### 12.2.2 Serum Chemistry

Parameters include albumin, ALP, ALT, amylase, AST, blood urea nitrogen, calcium, calculated creatinine clearance, carbon dioxide, chloride, creatinine, creatinine kinase and subtypes, gamma-glutamyl transferase, globulin, glucose (non-fasting), high-density lipoprotein, lactate dehydrogenase, lipase, low-density lipoprotein, magnesium, phosphorus, potassium, sodium, total bilirubin, direct bilirubin, total cholesterol, total protein, triglycerides and uric acid. Visits include EOS Visit RB-US-13-0003 and Day 169 Week 25 (EOS INDV-6000-301)/ET visit.

#### 12.2.3 Urinalysis

Parameters include appearance, bilirubin, color, glucose, ketones, leucocyte esterase, nitrite, occult blood, pH, protein, specific gravity and urobilinogen.

Microscopic examination of sediment will be performed only if the results of the urinalysis evaluation are positive. Microscopic examination also includes but not limited to WBC count, RBC count, casts, and crystals. The microscopic results will be listed only.

#### 12.3 VITAL SIGNS

Measurements of vital signs (supine blood pressure systolic, supine blood pressure diastolic, pulse rate, oral temperature, respiratory rate, pulse oximetry, weight, height, BMI, hip circumference, waist circumference and waist-to-hip ratio) will be summarized using descriptive statistics at each scheduled visit and time point including change from baseline, percentage change from baseline and pre- and post- injection change if available.

Listings/tables of all vital sign assessments will be provided for the following groups:

- Supine blood pressure systolic, Supine blood pressure diastolic, Pulse rate, Oral temperature, and Respiratory rate, Pulse Oximetry;
- Body weight, BMI, Hip Circumference, Waist Circumference and Waist-to-hip ratio.

#### 12.4 OTHER SAFETY PARAMETERS

#### 12.4.1 Suicidality

A listing of all results will be presented for all subjects for all visits.

Table summaries will be run twice with two different baseline definitions:

- "Baseline Lifetime" will use the answers for suicidality (lifetime) in the screening/baseline questionnaire.
- "Baseline 6 months" will use the answers for suicidality (in the past 6 months) in the screening/baseline questionnaire.

Suicidal Ideation Severity Scoring

RBP-6000 INDV-6000-301

Page 27

The suicidal ideation score ranges from 0 to 5 and depends on the answers to the suicidal ideation portion of the C-SSRS. The score is the maximum suicidal ideation category (in the following order: 1 = wish to be dead, 2 = non-specific active suicidal thoughts, 3 = active suicidal ideation with any methods (not plan) without intent to act, 4 = active suicidal ideation with some intent to act, without specific plan, and 5 = active suicidal ideation with specific plan and intent) present at the assessment. If none of these questions are YES, then the suicidal ideation score is 0.

#### Suicidal Ideation Intensity Scoring

The suicidal ideation intensity score is the sum of the five intensity item scores to create a total score (range 0 to 25). The five intensity items include frequency, duration, controllability, deterrents and reason for ideation. Each item is scored from 0 to 5 with 5 representing the most severe intensity.

#### Suicidal Behavior Scoring

The suicidal behavior score ranges from 0 to 5 and depends on the answers to the suicidal behavior portion of the C-SSRS. The score is the maximum suicidal behavior category (in the following order: 1 = preparatory acts or behavior, 2 = aborted attempt, 3 = interrupted attempt, 4 = actual attempt, and 5 if the subject has an AE with a preferred term of completed suicide. If none of these questions are YES and the subject does not have an AE with a preferred term of completed suicide, then the suicidal behavior score is 0.

Suicidal ideation and suicidal behavior responses (Yes/No) will be summarized by analysis visit using counts and percentages in the Safety Analysis Set. Shift tables to demonstrate changes in C-SSRS categories and changes in suicidal ideation and behavior scores from baseline during the Treatment Period will be presented. CSSRS and suicidal ideation responses will be listed separately. The suicidal ideation intensity ratings, each of the five items and the total score of the intensity for subjects with an ideation will be listed.

#### 12.4.2 Local Injection Site Evaluation

The local injection site will be evaluated for potential reaction and evidence of any attempts by the subject to remove RBP-6000 following a previous injection. A summary table and a listing will be provided. Attempted removal results will be summarized by percentage of subjects with attempted removal in each dose received at each visit.

#### 12.4.3 Local Injection Site Tolerability

Local injection site tolerability as assessed by the Injection Site Grading scale will be summarized and plotted over time by category (pain, tenderness, erythema/redness, induration, and swelling) and severity using frequency counts and percentages. Local injection site tolerability will be assigned a severity grade, including none (grade 0), mild (grade 1), moderate (grade 2), severe (grade 3), or potentially life threatening (grade 4) utilizing the 5-point Injection Site Grading Scale. A listing will be provided.

A separate listing will be presented for severe/life threatening responses with their corresponding VAS scores.

#### 12.4.4 Injection Site Pain

Injection Site Pain VAS scores will be summarized over time during the Treatment Period. And the maximum score during the Treatment Period will be calculated and tabulated. The burning/stinging categorical variable (Yes/No) will be summarized by percentage of responses in each dose received at each time point.

The percentage of subjects who reported injection site reaction (Yes) at each injection visit in the Safety Analysis Set. Mean value of local injection site VAS pain scores will also be plotted at each injection.

Separate listings for burning/stinging will be provided. A listing of injection site pain VAS scores will also be provided.

#### 12.4.5 Other Safety Variables

NA.

# 12.5 INDEPENDENT DRUG COUNSELING/BEHAVIOURAL THERAPY

A listing for whether independent drug counseling (IDC) was completed per subject visit will be provided.

# 13.0 POOLED ANALYSES

No pooled analyses will be conducted in this trial.

# **<u>14.0</u> <u>SUBGROUP ANALYSES</u>**

No subgroup analyses will be conducted in this trial.

# 15.0 HEALTH OUTCOME ANALYSES

No health outcome assessments were performed in this study.

# 16.0 PLASMA CONCENTRATION ANALYSES

No plasma concentration samples were collected in this study.

# 17.0 INTERIM ANALYSIS

No Interim analysis was performed for this study
# 18.0 DETERMINATION OF SAMPLE SIZE

This study is designed to provide ongoing treatment with RBP-6000 and to assess the safety monitoring for subjects who complete the RB-US-13-0003 study and for whom a new treatment venue has not been identified or arranged. Approximately 300 subjects who completed Study RB-US-13-0003 will be enrolled into this study.

# 19.0 COMPUTER METHODS

Statistical analyses will be performed using version 9.4 (or newer) of SAS on a Windows operating system.

### 20.0 DATA HANDLING CONVENTIONS

#### 20.1 REFERENCE DATES AND ANALYSIS PERIODS

There are two analysis periods in this study:

- Treatment Period (TP)
- Safety Follow-Up Period (SFU).

Treatment Period starts from Treatment Start Date and ends at Treatment End Date. Treatment Start Date (or Day 1) for a subject is the date of the first injection. Treatment End Date for a subject is the maximum of the date of the end-of-study/ Early Termination (EOS/ET) visit and the date of last injection + 28.

Safety Follow-Up Period starts from Safety Follow-Up Start Date and ends at Safety Follow-Up End Date, which are defined for all subject who have assessments in the Follow-Up period.

Safety Follow-Up Start Date for a subject is Treatment End Date +1.

Safety Follow-Up End Date for a subject is defined as the date of visit at Week 29 or unscheduled visit after the Treatment End Date (defined as above) for AE/concomitant medication reporting or lab/vital signs assessment, whichever comes later. That is, Follow-up end date is max (Follow-up Start Date, date of visit at Week 29, last unscheduled visit after the Treatment End Date to report AE/concomitant medication or to do lab/vital signs assessment, if available).

Any records collected prior to first injection date/time will be considered as Screening records. And any records collected after the Treatment End Date will be considered as Safety Follow-up records.

#### 20.2 ANALYSIS VISITS AND OTHER DEFINITIONS

All data will be presented in listings (including unscheduled visits), however only perprotocol visits will be summarized in tables and figures. Unscheduled and scheduled assessments will be utilized in the summaries for "at any time".

For lab values, body weight, BMI, waist circumference, hip circumference and waist-to-hip ratio, Early Termination and End-of-study results will be reported with the EOS/ET visit.

For all other assessments, occurring at the ET visit, will be mapped to the next perprotocol visit (or time point), that has not already been completed by the subject. A ET visit must not be mapped to a visit that a subject has already completed. RBP-6000 INDV-6000-301

V-6000-301 Page 37

The closest assessment value on or before Treatment Start Date/Time will be assigned as Baseline value and then be labeled as 'Baseline' in visit window, and for assessment prior to Treatment Start Date/Time, if exists, will be labeled as 'EOS 0003' or 'Screening' per its collecting time and per SOE definition.

For subjects who have one visit-based assessment in the Safety Follow-up (SFU) period, the period of the visit will be labeled as 'Safety Follow-Up Week 29'.

### **Other Definitions:**

#### **Subgroups**

#### Sex

- Male
- Female

#### **Age Categories**

- $\geq 18 \text{ to} < 30$
- $\geq 30 \text{ to} < 45$
- $\geq 45 \text{ to} < 60$
- ≥ 60
- ≥65

#### Race

- White
- Non-White

#### **Baseline BMI Categories**

- Under weight:  $0 \text{ to} < 18.5 \text{ kg/m}^2$
- Normal:  $\geq 18.5 \text{ kg/m}^2 \text{ and } \leq 25 \text{ kg/m}^2$
- Over weight:  $\geq 25 \text{ kg/m}^2 \text{ and } < 30 \text{ kg/m}^2$
- Obese:  $\geq 30 \text{ kg/m}^2$

#### **DERIVED EFFICACY VARIABLES** 20.3

Not applicable.

#### 20.4 REPEATED OR UNSCHEDULED ASSESSMENTS OF SAFETY **PARAMETERS**

See reference rules on unscheduled assessments in Section 20.2. Unscheduled assessments will be utilized in analyses "at any time" and will be listed in listings.

If there are more one assessments on one parameter at scheduled visits, the last assessment will be used for visit-based table/figure summaries.

#### 20.5 MISSING DATE OF INVESTIGATIONAL PRODUCT

When the date of the last injection of RBP-6000 during the Treatment Period is missing for a subject in the Safety Population, all efforts should be made to obtain the date from the investigator. If it is still missing after all efforts, then the last available dosing record date will be used as the last dose date.

#### 20.6 MISSING SEVERITY AND RELATIONSHIP TO STUDY DRUG IN ADVERSE EVENTS

If the severity is missing for an AE started on or after the date of the first dose of the investigational product, then a severity of "Severe" will be assigned.

If the relationship is missing for an AE started on or after the date of the first dose of the investigational product, then a relationship of "Related" will be assigned.

The imputed values for assessment will be used for incidence summary, while the actual values will be presented in data listings.

#### MISSING DATE INFORMATION FOR ADVERSE EVENTS 20.7

When the AE start date is incomplete (i.e., partially missing), then the following rules will be applied:

#### Missing day and month

- If the year is the same as the year of the date of the first dose of investigational product, then the day and month of the date of the first dose of investigational product will be assigned to the missing fields.
- If the year is before the year of the date of the first dose of investigational product, then December 31 will be assigned to the missing fields.


• If the year is after the year of the date of the first dose of investigational product, then January 1 will be assigned to the missing fields.

### Missing month only

• The day will be treated as missing and both month and day will be replaced according to the above procedure.

#### Missing day only

- If the month and year are the same as the month and year of the date of the first dose of investigational product, then the day of the first dose of investigational product will be assigned to the missing day.
- If either the year is before the year of the date of the first dose of investigational product or if both years are the same but the month is before the month of the date of the first dose of investigational product, then the last day of the month will be assigned to the missing day.
- If either the year is after the year of the date of the first dose of investigational product or if both years are the same but the month is after the month of the date of the first dose of investigational product, then the first day of the month will be assigned to the missing day.

If the stop date is after the date of the first dose of investigational product, the date of the first dose of investigational product will be assigned to the missing start date

If the stop date is before the date of the first dose of investigational product, the stop date will be assigned to the missing start date

# 20.8 MISSING DATE INFORMATION FOR CONCOMITANT MEDICATIONS

For concomitant medications, incomplete (i.e., partial missing) start date and/or stop date will be imputed. When the start date and the stop date are both incomplete for a subject, consider to impute the start date first.

#### Missing day and month

- If the year of the incomplete start date is the same as the year of the date of the first dose of investigational product, then the day and month of the date of the first dose will be assigned to the missing fields.
- If the year of the incomplete start date is before the year of the date of the first dose of investigational product, then December 31 will be assigned to the missing fields.
- If the year of the incomplete start date is after the year of the date of the first dose of investigational product, then January 1 will be assigned to the missing fields.

V-6000-301 Page 40

#### Missing month only

• The day will be treated as missing and both month and day will be replaced according to the above procedure.

#### Missing day only

- If the month and year of the incomplete start date are the same as the month and year of the date of the first dose of investigational product, then the day of the first dose will be assigned to the missing day.
- If either the year is before the year of the date of the first dose of investigational product or if both years are the same but the month is before the month of the date of the first dose of investigational product, then the last day of the month will be assigned to the missing day.
- If either the year is after the year of the date of the first dose of investigational product or if both years are the same but the month is after the month of the date of the first dose of investigational product, then the first day of the month will be assigned to the missing day.

#### **Incomplete Stop Date**

#### Missing day and month

- If the year of the incomplete stop date is the same as the year of the date of the last dose of investigational product, then the day and month of the date of the last dose will be assigned to the missing fields.
- If the year of the incomplete stop date is before the year of the date of the last dose of investigational product, then December 31 will be assigned to the missing fields.
- If the year of the incomplete stop date is after the year of the date of the last dose of investigational product, then January 1 will be assigned to the missing fields.

#### Missing month only

• The day will be treated as missing and both month and day will be replaced according to the above procedure.

#### Missing day only

- If the month and year of the incomplete stop date are the same as the month and year of the date of the last dose of investigational product, then the day of the last dose will be assigned to the missing day.
- If either the year is before the year of the date of the last dose of investigational product or if both years are the same but the month is before the month of the date of the last dose of investigational product, then the last day of the month will be assigned to the missing day.

• If either the year is after the year of the date of the last dose of investigational product or if both years are the same but the month is after the month of the date of the last dose of investigational product, then the first day of the month will be assigned to the missing day.

# 20.9 CHARACTER VALUES OF CLINICAL LABORATORY PARAMETERS AND OTHER LABORATORY IMPUTATION RULES

- If a reported value of a clinical laboratory parameter cannot be used in a statistical summary table due, for example, to the fact that a character string is reported for a parameter of the numerical type, a coded value needs to be appropriately determined and used in the statistical analyses. Value of X+0.0001 will be used to impute ">X" character value and X-0.0001 will be used to impute "<X". That is, if X equal to 60, 60.0001 will be used to impute character value of ">60" and 59.999 will be used to impute "<60". However, the actual values as reported in the database may be presented in data listings.
- Due to the fact that screening lab records were rolled-over from RB-US-13-0003, whose LDH, total bilirubin and AST records have lower limits and HDL-C records have upper limit as opposed to at visits after first injection only having one-sided upper limits for parameters LDH, total bilirubin and AST and one-sided lower limit for HDL-C, lab classification values (i.e., Low, normal and high) for parameters LDH, total bilirubin and AST and HDL-C at screening and from RB-US-13-0003 should be imputed so that shift tables can be tabulated. The imputation rules are as follows:
  - o For screening records (ie, rolled-over from RB-US-13-0003) of parameters LDH, total bilirubin and AST, lower limits will be imputed as 0. The lab character values of "Low" and "Normal" will be collapsed to be "Normal".
  - For screening records (ie, rolled-over from RB-US-13-0003) of HDL-C, upper limit will be imputed as blank. The lab character values of "Normal" and "High" will be collapsed to be "Normal".
- GGT assessments at Screening have categories of normal and high but have three categories of low, normal and high post-baseline. Then for GGT post-baseline assessments, low and normal will be collapsed to normal.

#### 20.10 C-SSRS DATA IMPUTATION

In the Suicidal Behavior section, when the answer to the question "Have you made a suicide attemp" is NO, then the "Total # of Attempts" should be 0. In our clincial database, we have both 0 and Blank present. In the analysis dataset, under this scenario, Blank for Total # of Attempts will be imputed as 0.

# 21.0 CHANGES TO ANALYSES SPECIFIED IN PROTOCOL

No changes have been made to analyses specified in protocol.

# **<u>22.0</u> <u>REFERENCES</u>**

Guidance for Industry Drug-Induced Liver Injury: Premarketing Clinical Evaluation: U.S. Department of Health and Human Services Food and Drug Administration Center for Drug Evaluation and Research (CDER) Center for Biologics Evaluation and Research (CBER)

# 23.0 APPENDIX

# 23.1 APPENDIX 1: LIST OF PREFERRED TERMS FROM STANDARD MEDDRA QUERIES FOR ADVERSE EVENTS OF SPECIAL INTEREST

# LIST OF PREFERRED TERMS FOR PSYCHIATRIC HISTORY

| Adjustment disorder with anxiety | Cyclothymic disorder |
|---|---|
| Adjustment disorder with depressed mood | Bipolar disorder |
| Adjustment disorder with disturbance of | |
| conduct | Hypomania |
| Adjustment disorder with mixed anxiety | |
| and depressed mood | Mania |
| Adjustment disorder with mixed disturbance of emotion and conduct | Diviste d officet |
| | Blunted affect |
| Grief reaction | Constricted affect |
| Adjustment disorder | Flat affect |
| Agitation | Inappropriate affect |
| Agitation neonatal | Affect lability |
| Anticipatory anxiety | Affective ambivalence |
| Anxiety | Anger |
| Nervousness | Dysphoria |
| Stress | Emotional disorder |
| Tension | Emotional poverty |
| Activation syndrome | Euphoric mood |
| Acute stress disorder | Irritability |
| Post-traumatic stress disorder | Moaning |
| Postpartum stress disorder | Mood altered |
| Burnout syndrome | Emotional distress |
| Anniversary reaction | Neuroleptic-induced deficit syndrome |
| Acrophobia | Alexithymia |
| Agoraphobia | Frustration tolerance decreased |
| Animal phobia | Mood swings |
| Claustrophobia | Affective disorder |
| Fear | Apathy |
| Fear of animals | Listless |
| Fear of closed spaces | Mood disorder due to a general medical condition |
| Fear of disease | Seasonal affective disorder |
| Fear of open spaces | Boredom |

|------------------------------|-------------------------------------------|
| Fear of weight gain | Laziness |
| Performance fear | Substance-induced mood disorder |
| Phobia | Aggression |
| Phobia of exams | Antisocial behaviour |
| Phobia of flying | Asocial behaviour |
| Phobic avoidance | Attention-seeking behaviour |
| Social anxiety disorder | Belligerence |
| Social fear | Disinhibition |
| Fear of falling | Grandiosity |
| Dysmorphophobia | Hostility |
| Ochlophobia | Indifference |
| Phagophobia | Inferiority complex |
| Fear of crowded places | Negativism |
| Fear of eating | Paranoia |
| Arachnophobia | Personality change |
| Hydrophobia | Social avoidant behaviour |
| Phonophobia | Soliloquy |
| Phobia of driving | Suspiciousness |
| Noctiphobia | Violence-related symptom |
| Nocturnal fear | Homicidal ideation |
| Osmophobia | Impatience |
| Nosophobia | Disturbance in social behaviour |
| Photaugiaphobia | Aversion |
| Thanatophobia | Suggestibility |
| Fear of death | Stubbornness |
| Fear of pregnancy | Pseudologia |
| Haphephobia | Overconfidence |
| Paruresis | Egocentrism |
| Pharmacophobia | Defiant behaviour |
| Emetophobia | Personality disorder |
| Autophobia | Pithiatism |
| Haemophobia | Self esteem decreased |
| Fear of injection | Self esteem inflated |
| Thermophobia | Avoidant personality disorder |
| Algophobia | Dependent personality disorder |
| Limited symptom panic attack | Obsessive-compulsive personality disorder |
| Panic attack | Antisocial personality disorder |
| Panic disorder | Borderline personality disorder |
| Panic reaction | Histrionic personality disorder |

| Compulsions | Narcissistic personality disorder |
|---|---|
| Obsessive thoughts | Psychopathic personality |
| Obsessive-compulsive disorder | Paranoid personality disorder |
| Trichotillomania | Schizoid personality disorder |
| Body dysmorphic disorder | Schizotypal personality disorder |
| Obsessive rumination | Breath holding |
| Dermatillomania | Staring |
| Compulsive lip biting | Regressive behaviour |
| Nail picking | Abnormal behaviour |
| Compulsive shopping | Sexually inappropriate behaviour |
| Compulsive hoarding | Behaviour disorder due to a general medical condition |
| Compulsive handwashing | Scatolia |
| Paediatric autoimmune neuropsychiatric | |
| disorders associated with streptococcal | |
| infection | Neglect of personal appearance |
| Trichotemnomania | Trance |
| Compulsive cheek biting | Hypervigilance |
| Obsessive need for symmetry | Abulia |
| Obsessive-compulsive symptom | Psychiatric symptom |
| Anxiety disorder due to a general medical | |
| condition | Psychiatric decompensation |
| Generalised anxiety disorder | Decreased eye contact |
| Neurosis | Psychological trauma |
| Postpartum neurosis | Helplessness |
| Selective mutism | Personality change due to a general medical condition |
| Separation anxiety disorder | Mental disorder due to a general medical condition |
| Anxiety disorder | Neuropsychiatric syndrome |
| Catatonia | Psychological factor affecting medical condition |
| Restlessness | Mental status changes |
| Automatism | Dyslogia |
| Automatism epileptic | Mental disorder |
| Automatism, command | Emotional disorder of childhood |
| Bruxism | Neurotic disorder of childhood |
| Echolalia | Personality disorder of childhood |
| Ed | Reactive attachment disorder of infancy or early |
| Echopraxia | childhood |
| Head banging | School refusal |
| Posturing | Disinhibited social engagement disorder of childhood |
| Stereotypy | Encopresis |
| Waxy flexibility | Enuresis |

| 111/1/1-0000-301 | Tuge 47 |
|---|---|
| Tic | Alcohol abuse |
| Chronic tic disorder | Alcohol problem |
| Complex tic | Alcoholic hangover |
| Provisional tic disorder | Alcoholism |
| Secondary tic | Dependence |
| Attention deficit/hyperactivity disorder | Drug abuse |
| Atypical attention deficit syndrome | Drug dependence |
| Oppositional defiant disorder | Drug dependence, antepartum |
| Conduct disorder | Drug dependence, postpartum |
| Disruptive mood dysregulation disorder | Tobacco abuse |
| Change in sustained attention | Withdrawal syndrome |
| Distractibility | Alcohol withdrawal syndrome |
| Daydreaming | Nicotine dependence |
| Executive dysfunction | Tobacco withdrawal symptoms |
| Vascular cognitive impairment | Neonatal complications of substance abuse |
| Mental fatigue | Substance abuse |
| Learning disability | Dopamine dysregulation syndrome |
| Reading disorder | Binge drinking |
| Learning disorder | Substance dependence |
| Mutism | Gambling disorder |
| Communication disorder | Brief psychotic disorder, with postpartum onset |
| Speech sound disorder | Brief psychotic disorder with marked stressors |
| Clang associations | Transient psychosis |
| Logorrhoea | Brief psychotic disorder without marked stressors |
| Neologism | Alice in wonderland syndrome |
| Verbigeration | Delusional disorder, erotomanic type |
| Taciturnity | Delusional disorder, grandiose type |
| Disorganised speech | Delusional disorder, jealous type |
| Coprolalia | Delusional disorder, mixed type |
| Lack of spontaneous speech | Delusional disorder, somatic type |
| Poverty of speech | Delusional disorder, unspecified type |
| Pressure of speech | Delusional disorder, persecutory type |
| Screaming | Acute psychosis |
| Dysphemia | Alcoholic psychosis |
| Confusional state | Psychotic behaviour |
| Disorientation | Senile psychosis |
| Delirium | Shared psychotic disorder |
| Delirium tremens | Reactive psychosis |
| Delirium febrile | Epileptic psychosis |

| 11/1/27-0000-301 | Tuge 40 |
|---|---|
| Post-traumatic amnestic disorder | Childhood psychosis |
| Korsakoff's syndrome | Psychotic disorder |
| Paramnesia | Psychotic disorder due to a general medical condition |
| Pseudodementia | Hysterical psychosis |
| Behavioural and psychiatric symptoms of | |
| dementia | Postictal psychosis |
| Agitated depression | Substance-induced psychotic disorder |
| Depression | Rebound psychosis |
| Depression suicidal | Parkinson's disease psychosis |
| Postpartum depression | Schizoaffective disorder |
| Major depression | Schizophreniform disorder |
| Menopausal depression | Schizoaffective disorder bipolar type |
| Childhood depression | Schizoaffective disorder depressive type |
| Post stroke depression | Schizophrenia |
| Postictal depression | Anorgasmia |
| Persistent depressive disorder | Female orgasmic disorder |
| Anhedonia | Male orgasmic disorder |
| Decreased interest | Orgasm abnormal |
| Depressed mood | Premature ejaculation |
| Feeling of despair | Orgasmic sensation decreased |
| Feelings of worthlessness | Psychosexual disorder |
| Morose | Sex dysphoria |
| Psychomotor retardation | Sexual inhibition |
| Tearfulness | Psychogenic erectile dysfunction |
| Feeling guilty | Disturbance in sexual arousal |
| Depressive symptom | Excessive masturbation |
| Negative thoughts | Libido decreased |
| Sense of a foreshortened future | Libido increased |
| Autism spectrum disorder | Loss of libido |
| Neurodevelopmental disorder | Sexual aversion disorder |
| Dissociation | Excessive sexual fantasies |
| Dissociative amnesia | Libido disorder |
| Dissociative disorder | Hypersexuality |
| Dissociative identity disorder | Compulsive sexual behaviour |
| Depersonalisation/derealisation disorder | Genito-pelvic pain/penetration disorder |
| Delusion | Exhibitionism |
| Delusion of grandeur | Fetishism |
| Delusion of reference | Frotteurism |
| Delusion of replacement | Masochism |
| · | I . |

| 111/11/11/11/11 | 1 uge 47 |
|---|---|
| Erotomanic delusion | Paedophilia |
| Jealous delusion | Paraphilia |
| Persecutory delusion | Sadism |
| Somatic delusion | Transvestism |
| Thought insertion | Voyeurism |
| Thought withdrawal | Initial insomnia |
| Thought broadcasting | Insomnia |
| Cotard's syndrome | Middle insomnia |
| Depressive delusion | Hyposomnia |
| Mixed delusion | Terminal insomnia |
| Deja vu | Behavioural insomnia of childhood |
| Delusional perception | Breathing-related sleep disorder |
| Derealisation | Dyssomnia |
| Flashback | Hypnagogic hallucination |
| Hallucination | Hypnopompic hallucination |
| Hallucination, auditory | Sleep attacks |
| Hallucination, gustatory | Abnormal dreams |
| Hallucination, olfactory | Nightmare |
| Hallucination, tactile | Rapid eye movements sleep abnormal |
| Hallucination, visual | Sleep talking |
| Hallucinations, mixed | Sleep terror |
| Illusion | Somnambulism |
| Jamais vu | Abnormal sleep-related event |
| Somatic hallucination | Parasomnia |
| Hallucination, synaesthetic | Loss of dreaming |
| Paroxysmal perceptual alteration | Sleep-related eating disorder |
| Time perception altered | Sleep sex |
| Autoscopy | Sleep inertia |
| Circumstantiality | Confusional arousal |
| Confabulation | Rapid eye movement sleep behaviour disorder |
| | Sleep disorder due to general medical condition, |
| Derailment | hypersomnia type |
| 51: 1 : 6: 1 | Sleep disorder due to general medical condition, |
| Flight of ideas | insomnia type |
| Ideas of reference | Sleep disorder due to general medical condition, mixed type |
| Tacas of reference | Sleep disorder due to general medical condition, |
| Illogical thinking | parasomnia type |
| Loose associations | Sleep disorder due to a general medical condition |
| Magical thinking | Sleep disorder |
| | 1 1 |

| | - 1.81 1 % |
|---|---|
| Perseveration | Hypersomnia-bulimia syndrome |
| Poverty of thought content | Sopor |
| Tangentiality | Hypersomnia related to another mental condition |
| Thinking abnormal | Insomnia related to another mental condition |
| Thought blocking | Completed suicide |
| Bradyphrenia | Intentional self-injury |
| Morbid thoughts | Suicidal ideation |
| Intellectualisation | Suicide attempt |
| Tachyphrenia | Self-injurious ideation |
| Impaired reasoning | Self injurious behaviour |
| Paralogism | Suicidal behaviour |
| Pathological doubt | Suicide threat |
| Intrusive thoughts | Compensation neurosis |
| Purging | Munchausen's syndrome |
| Self-induced vomiting | Factitious disorder |
| Eating disorder symptom | Conversion disorder |
| Anorexia and bulimia syndrome | Polydipsia psychogenic |
| Anorexia nervosa | Psychogenic dysuria |
| Binge eating | Torticollis psychogenic |
| Bulimia nervosa | Vomiting psychogenic |
| Eating disorder | Psychosomatic disease |
| Merycism | Pseudoneurologic symptom |
| Pica | Psychogenic seizure |
| Food aversion | Psychogenic movement disorder |
| Selective eating disorder | Psychogenic tremor |
| Impulsive behaviour | Psychogenic respiratory distress |
| Intermittent explosive disorder | Somatoform genitourinary disorder |
| Kleptomania | Somatic symptom disorder |
| Poriomania | Illness anxiety disorder |
| Pyromania | Cardiovascular somatic symptom disorder |
| Onychophagia | Gastrointestinal somatic symptom disorder |
| Impulse-control disorder | Neurologic somatic symptom disorder |
| Necromania | Cutaneous somatic symptom disorder |
| Clinomania | Somatic symptom disorder of pregnancy |
| Bipolar I disorder | |
| Bipolar II disorder | |

# CUSTOMIZED MEDDRA QUERY (CMQ) LIST OF PREFERRED TERMS FOR DRUG RELATED HEPATIC DISORDERS

| Cholestasis and jaundice of hepatic or | igin |
|---|---|
| Bilirubin excretion disorder | Jaundice |
| Cholaemia | Jaundice cholestatic |
| Cholestasis | Jaundice hepatocellular |
| Cholestatic liver injury | Mixed liver injury |
| Cholestatic pruritus | Ocular icterus |
| Drug-induced liver injury | Parenteral nutrition associated liver disease |
| Hepatitis cholestatic | Deficiency of bile secretion |
| Hyperbilirubinaemia | Yellow skin |
| Icterus index increased | |
| Hepatic failure, fibrosis and cirrhosis | and other liver damage-related conditions |
| Acute hepatic failure | Liver and small intestine transplant |
| Acute on chronic liver failure | Liver dialysis |
| Acute yellow liver atrophy | Liver disorder |
| Ascites | Liver injury |
| Asterixis | Liver operation |
| Bacterascites | Liver transplant |
| Biliary cirrhosis | Lupoid hepatic cirrhosis |
| Biliary cirrhosis primary | Minimal hepatic encephalopathy |
| Biliary fibrosis | Mixed liver injury |
| Cholestatic liver injury | Nodular regenerative hyperplasia |
| Chronic hepatic failure | Non-alcoholic fatty liver |
| Coma hepatic | Non-alcoholic steatohepatitis |
| Cryptogenic cirrhosis | Non-cirrhotic portal hypertension |
| Diabetic hepatopathy | Oedema due to hepatic disease |
| Drug-induced liver injury | Oesophageal varices haemorrhage |
| Duodenal varices | Peripancreatic varices |
| Gallbladder varices | Portal fibrosis |
| Gastric variceal injection | Portal hypertension |
| Gastric variceal ligation | Portal hypertensive enteropathy |
| Gastric varices | Portal hypertensive gastropathy |
| Gastric varices haemorrhage | Portal vein cavernous transformation |

| Hepatic atrophy Portal vein dilatation Hepatic atrophy Porto pulmonary hypertension Hepatic calcification Renal and liver transplant Hepatic cirrhosis Retrograde portal vein flow Hepatic encephalopathy Reye's syndrome Hepatic encephalopathy prophylaxis Reynold's syndrome Hepatic failure Splenic varices Hepatic fibrosis Splenic varices Hepatic infiltration eosinophilic Subacute hepatitis Hepatic infiltration eosinophilic Subacute hepatic failure Hepatic lesion Varices oesophageal Hepatic seatosis Varicose veins of abdominal wall Hepatic steato-fibrosis Anorectal varices Hepatitis fulminant Intrahepatic portal hepatic venous fistula Hepatobiliary disease Peritoneovenous shunt Hepatocellular foamy cell syndrome Portal shunt Hepatocellular injury Portal shunt procedure Hepatorenal failure Spider naevus Hepatorenal failure Spider naevus Hepatoronal failure Spider naevus Hepatoroxicity Splenorenal shunt procedure Intestinal varices haemorrhage Stomal varices Varicose vein Hepatitis, non-infectious Acute graft versus host disease in liver Hepatitis fulminant Hepatitis fulminant Hepatitis fulminant Hepatitis fulminant Intestinal varices haemorrhage Stomal varices Varicose vein Hepatitis on-infectious Acute graft versus host disease in liver Hepatitis fulminant | 111/1/27-0000-301 | |
|---|---|---|
| Hepatic calcification Renal and liver transplant Hepatic cirrhosis Retrograde portal vein flow Hepatic encephalopathy Reye's syndrome Hepatic encephalopathy prophylaxis Reynold's syndrome Hepatic failure Splenic varices Hepatic fibrosis Splenic varices haemorrhage Hepatic hydrothorax Steatohepatitis Hepatic lesion Varices oesophageal Hepatic lesion Varices oesophageal Hepatic steato-fibrosis Anorectal varices Hepatic steato-fibrosis Anorectal varices haemorrhage Hepatitis fulminant Intrahepatic portal shunt Pepatocellular foamy cell syndrome Hepatocellular foamy cell syndrome Portal shunt procedure Hepatorenal failure Spider naevus Hepatorenal syndrome Splenorenal shunt Hepatotoxicity Splenorenal shunt procedure Varicose vein Hepatitis, non-infectious Acute graft versus host disease in liver Allergic hepatitis Hepatitis (hepatitis Chronic graft versus host disease in liver Radiation hepatitis Hepatitis Steatohepatitis Steatohepatitis Hepatitis ohlestatic Liver sarcoidosis | Hepatectomy | Portal vein dilatation |
| Hepatic cirrhosis Retrograde portal vein flow Hepatic encephalopathy Reye's syndrome Hepatic encephalopathy prophylaxis Reynold's syndrome Hepatic failure Splenic varices Hepatic fibrosis Splenic varices haemorrhage Hepatic hydrothorax Steatohepatitis Hepatic lesion Varices oesophageal Hepatic lesion Varices oesophageal Hepatic steato-fibrosis Anorectal varices Hepatic steatosis Anorectal varices Hepatitis fulminant Intrahepatic portal hepatic venous fistula Hepatosuclellular foamy cell syndrome Portal shunt Hepatocellular injury Portal shunt Hepatocellular injury Portal shunt procedure Hepatorenal failure Spider naevus Hepatorenal syndrome Splenorenal shunt Hepatoroxicity Splenorenal shunt procedure Intestinal varices haemorrhage Stomal varices Varicose vein Hepatitis fulminant Hepatitis, non-infectious Acute graft versus host disease in liver Allergic hepatitis Chronic graft versus host disease in liver Radiation hepatitis Hepatitis Steatohepatitis Steatohepatitis Hepatitis Steatohepatitis Hepatitis Acute Granulomatous liver disease Hepatitis cholestatic Liver sarcoidosis | Hepatic atrophy | Porto pulmonary hypertension |
| Hepatic encephalopathy Reye's syndrome Hepatic encephalopathy prophylaxis Reynold's syndrome Hepatic failure Splenic varices Hepatic fibrosis Splenic varices haemorrhage Hepatic infiltration eosinophilic Subacute hepatic failure Hepatic infiltration eosinophilic Subacute hepatic failure Hepatic lesion Varices oesophageal Hepatic necrosis Varicose veins of abdominal wall Hepatic steato-fibrosis Anorectal varices Hepatic steatosis Anorectal varices Hepatic steatosis Anorectal varices haemorrhage Hepatitis fulminant Intrahepatic portal hepatic venous fistula Hepatocellular foamy cell syndrome Portal shunt procedure Hepatocellular injury Portal shunt procedure Hepatopulmonary syndrome Small-for-size liver syndrome Hepatorenal failure Splenorenal shunt Hepatorenal syndrome Splenorenal shunt Hepatorenal syndrome Splenorenal shunt Hepatorenal varices Spontaneous intrahepatic portosystemic venous shunt Intestinal varices haemorrhage Stomal varices Varicose vein Hepatitis fulminant Allergic hepatitis Hepatitis fulminant Allergic hepatitis Hepatitis fulminant Allergic hepatitis Hepatitis fulminant Chronic graft versus host disease in liver Lupus hepatitis Chronic graft versus host disease in liver Radiation hepatitis Graft versus host disease in liver Radiation hepatitis Hepatitis Acute Granulomatous liver disease Hepatitis coute Liver sarcoidosis | Hepatic calcification | Renal and liver transplant |
| Hepatic encephalopathy prophylaxis Hepatic failure Splenic varices Subacute hepatic failure Warices oesophageal Warices oesophageal Warices oesophageal Warices veins of abdominal wall Warices oesophageal Warices veins of abdominal wall Warices oesophageal Warices veins of abdominal wall Warices oesophageal Warices veins of abdominal wall Warices veins of abdominal wall Warices oensor fabdominal wall Wari | Hepatic cirrhosis | Retrograde portal vein flow |
| Hepatic failure Hepatic fibrosis Splenic varices Splenic varices haemorrhage Hepatic hydrothorax Steatohepatitis Hepatic infiltration eosinophilic Hepatic lesion Hepatic lesion Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steatosis Hepatic steatosis Hepatitis fulminant Hepatobiliary disease Hepatocellular foamy cell syndrome Hepatocellular injury Portal shunt Hepatopulmonary syndrome Hepatorenal failure Spider naevus Hepatoroxicity Intestinal varices Spontaneous intrahepatic portosystemic venous shunt Intestinal varices Varicose vein Hepatitis, non-infectious Acute graft versus host disease in liver Allergic hepatitis Chronic graft versus host disease in liver Hepatitis Hepatitis cute Hepatitis cute Granulomatous liver disease Liver sarcoidosis | Hepatic encephalopathy | Reye's syndrome |
| Hepatic fibrosis Hepatic hydrothorax Hepatic infiltration eosinophilic Hepatic lesion Hepatic lesion Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steatosis Hepatic steatosis Hepatic steatosis Hepatic steatobiliary disease Hepatocellular foamy cell syndrome Hepatocullular injury Hepatopulmonary syndrome Hepatorenal failure Hepatorenal failure Hepatoxicity Intestinal varices Non-alcoholic steatosi Acute graft versus host disease in liver Chronic graft versus host disease in liver Hepatitis fulminant Hepatitis fulminant Hepatitis fulminant Hepatocellular foamy cell syndrome Portal shunt procedure Portal shunt procedure Small-for-size liver syndrome Splenorenal shunt Splenorenal shunt Splenorenal shunt Splenorenal shunt Foredure Spontaneous intrahepatic portosystemic venous shunt Hepatitis, non-infectious Acute graft versus host disease in liver Hepatitis Chronic graft versus host disease in liver Chronic hepatitis Foraft versus host disease in liver Hepatitis Foraft versus host disease in liver Hepatitis Foraft versus host disease in liver Hepatitis Foraft versus host disease in liver Radiation hepatitis Hepatitis acute Hepatitis coute Liver sarcoidosis | Hepatic encephalopathy prophylaxis | Reynold's syndrome |
| Hepatic hydrothorax Hepatic infiltration eosinophilic Hepatic lesion Varices oesophageal Hepatic steato-fibrosis Hepatic steato-fibrosis Hepatic steatosis Hepatic steatosis Hepatic steatosis Hepatic steatobiliary disease Hepatocellular foamy cell syndrome Hepatopulmonary syndrome Hepatopulmonary syndrome Hepatorenal failure Hepatotoxicity Intestinal varices Acute graft versus host disease in liver Allergic hepatitis Chronic graft versus host disease in liver Hepatitis fulminant Hepatoboliary disease Peritoneovenous shunt Hepatocellular foamy cell syndrome Portal shunt Portal shunt Portal shunt Procedure Small-for-size liver syndrome Spiden naevus Splenorenal shunt Splenorenal shunt Splenorenal shunt Splenorenal shunt Foredure Spontaneous intrahepatic portosystemic venous shunt Intestinal varices Hepatitis, non-infectious Acute graft versus host disease in liver Allergic hepatitis Autoimmune hepatitis Chronic graft versus host disease in liver Chronic hepatitis Chronic hepatitis Foraft versus host disease in liver Hepatitis cute Hepatitis cute Hepatitis cute Hepatitis cute Granulomatous liver disease Liver sarcoidosis | Hepatic failure | Splenic varices |
| Hepatic infiltration eosinophilic Hepatic lesion Varices oesophageal Varicose veins of abdominal wall Hepatic steato-fibrosis Anorectal varices Hepatic steatosis Anorectal varices haemorrhage Hepatitis fulminant Hepatobiliary disease Peritoneovenous shunt Hepatocellular foamy cell syndrome Hepatocellular injury Portal shunt procedure Hepatopulmonary syndrome Small-for-size liver syndrome Hepatorenal failure Spider naevus Hepatorenal syndrome Splenorenal shunt Hepatotoxicity Splenorenal shunt procedure Intestinal varices Spontaneous intrahepatic portosystemic venous shunt Intestinal varices haemorrhage Stomal varices Varicose vein Hepatitis, non-infectious Acute graft versus host disease in liver Allergic hepatitis Autoimmune hepatitis Chronic graft versus host disease in liver Chronic hepatitis Non-alcoholic steatohepatitis Graft versus host disease in liver Radiation hepatitis Hepatitis acute Hepatitis cholestatic Liver sarcoidosis | Hepatic fibrosis | Splenic varices haemorrhage |
| Hepatic lesion Varices oesophageal Hepatic necrosis Varicose veins of abdominal wall Hepatic steato-fibrosis Anorectal varices Hepatic steatosis Anorectal varices haemorrhage Hepatitis fulminant Intrahepatic portal hepatic venous fistula Hepatobiliary disease Peritoneovenous shunt Hepatocellular foamy cell syndrome Portal shunt procedure Hepatopulmonary syndrome Small-for-size liver syndrome Hepatorenal failure Spider naevus Hepatorenal syndrome Splenorenal shunt Hepatotoxicity Splenorenal shunt procedure Intestinal varices Spontaneous intrahepatic portosystemic venous shunt Intestinal varices haemorrhage Stomal varices Varicose vein Hepatitis, non-infectious Acute graft versus host disease in liver Hepatitis fulminant Allergic hepatitis Hepatitis Chronic graft versus host disease in liver Lupus hepatitis Chronic fepatitis Non-alcoholic steatohepatitis Graft versus host disease in liver Radiation hepatitis Hepatitis acute Hepatitis cholestatic Liver sarcoidosis | Hepatic hydrothorax | Steatohepatitis |
| Hepatic necrosis Hepatic steato-fibrosis Hepatic steatosis Hepatic steatosis Hepatitis fulminant Hepatitis fulminant Hepatobiliary disease Hepatocellular foamy cell syndrome Hepatocellular injury Hepatopulmonary syndrome Hepatorenal failure Hepatorenal syndrome Hepatorenal syndrome Hepatorenal syndrome Spider naevus Splenorenal shunt Hepatotoxicity Intestinal varices Spontaneous intrahepatic portosystemic venous fistula Hepatitis, non-infectious Acute graft versus host disease in liver Allergic hepatitis Chronic graft versus host disease in liver Chronic hepatitis Graft versus host disease in liver Hepatitis acute Hepatitis cholestatic Liver sarcoidosis Liver sarcoidosis | Hepatic infiltration eosinophilic | Subacute hepatic failure |
| Hepatic steato-fibrosis Hepatic steatosis Anorectal varices haemorrhage Hepatitis fulminant Hepatobiliary disease Hepatocellular foamy cell syndrome Hepatocellular injury Portal shunt procedure Hepatorenal failure Hepatorenal syndrome Hepatotoxicity Intestinal varices haemorrhage Varicose vein Hepatitis Acute graft versus host disease in liver Chronic graft versus host disease in liver Hepatitis Graft versus host disease in liver Hepatitis acute Hepatitis cholestatic Granulomatous liver disease Hepatitis cholestatic Liver sarcoidosis | Hepatic lesion | Varices oesophageal |
| Hepatitis fulminant Intrahepatic portal hepatic venous fistula Hepatobiliary disease Peritoneovenous shunt Hepatocellular foamy cell syndrome Portal shunt procedure Hepatopulmonary syndrome Small-for-size liver syndrome Hepatorenal failure Spider naevus Hepatorenal syndrome Splenorenal shunt Hepatotoxicity Splenorenal shunt procedure Intestinal varices Spontaneous intrahepatic portosystemic venous shunt Intestinal varices haemorrhage Stomal varices Varicose vein Hepatitis, non-infectious Acute graft versus host disease in liver Hepatitis fulminant Allergic hepatitis Hepatitis Chronic graft versus host disease in liver Lupus hepatitis Chronic graft versus host disease in liver Radiation hepatitis Graft versus host disease in liver Radiation hepatitis Hepatitis acute Granulomatous liver disease Hepatitis cholestatic Liver sarcoidosis | Hepatic necrosis | Varicose veins of abdominal wall |
| Hepatitis fulminant Intrahepatic portal hepatic venous fistula Hepatobiliary disease Peritoneovenous shunt Hepatocellular foamy cell syndrome Portal shunt Hepatocellular injury Portal shunt procedure Hepatopulmonary syndrome Small-for-size liver syndrome Hepatorenal failure Spider naevus Hepatorenal syndrome Splenorenal shunt Hepatotoxicity Splenorenal shunt procedure Intestinal varices Spontaneous intrahepatic portosystemic venous shunt Intestinal varices haemorrhage Stomal varices Varicose vein Hepatitis, non-infectious Acute graft versus host disease in liver Hepatitis fulminant Allergic hepatitis Hepatitis Chronic graft versus host disease in liver Lupus hepatitis Chronic praft versus host disease in liver Lupus hepatitis Chronic hepatitis Non-alcoholic steatohepatitis Graft versus host disease in liver Radiation hepatitis Hepatitis Steatohepatitis Hepatitis acute Granulomatous liver disease Liver sarcoidosis | Hepatic steato-fibrosis | Anorectal varices |
| Hepatocellular foamy cell syndrome Portal shunt Hepatocellular injury Portal shunt procedure Hepatopulmonary syndrome Hepatorenal failure Spider naevus Hepatorenal syndrome Splenorenal shunt Hepatotoxicity Splenorenal shunt procedure Intestinal varices Spontaneous intrahepatic portosystemic venous shunt Intestinal varices haemorrhage Varicose vein Hepatitis, non-infectious Acute graft versus host disease in liver Allergic hepatitis Chronic graft versus host disease in liver Chronic hepatitis Graft versus host disease in liver Hepatitis Hepatitis Graft versus host disease in liver Hepatitis Hepatitis Lupus hepatitis Graft versus host disease in liver Radiation hepatitis Hepatitis Hepatitis acute Granulomatous liver disease Hepatitis cholestatic Liver sarcoidosis | Hepatic steatosis | Anorectal varices haemorrhage |
| Hepatocellular foamy cell syndrome Portal shunt Hepatocellular injury Portal shunt procedure Hepatopulmonary syndrome Small-for-size liver syndrome Hepatorenal failure Spider naevus Hepatorenal syndrome Splenorenal shunt Hepatotoxicity Splenorenal shunt procedure Intestinal varices Spontaneous intrahepatic portosystemic venous shunt Intestinal varices haemorrhage Stomal varices Varicose vein Hepatitis, non-infectious Acute graft versus host disease in liver Allergic hepatitis Hepatitis toxic Autoimmune hepatitis Chronic graft versus host disease in liver Chronic hepatitis Chronic hepatitis Graft versus host disease in liver Radiation hepatitis Hepatitis acute Hepatitis cholestatic Liver sarcoidosis | Hepatitis fulminant | Intrahepatic portal hepatic venous fistula |
| Hepatocellular injury Portal shunt procedure Hepatopulmonary syndrome Small-for-size liver syndrome Hepatorenal failure Spider naevus Hepatorenal syndrome Splenorenal shunt Hepatotoxicity Splenorenal shunt procedure Intestinal varices Spontaneous intrahepatic portosystemic venous shunt Intestinal varices haemorrhage Varicose vein Hepatitis, non-infectious Acute graft versus host disease in liver Allergic hepatitis Hepatitis toxic Autoimmune hepatitis Chronic graft versus host disease in liver Chronic hepatitis Foraft versus host disease in liver Hepatitis Foraft versus host disease in liver Hepatitis Foraft versus host disease in liver Hepatitis Foraft versus host disease in liver Hepatitis Foraft versus host disease in liver Hepatitis Hepatitis Foraft versus host disease in liver Hepatitis Hepatitis Liver sarcoidosis | Hepatobiliary disease | Peritoneovenous shunt |
| Hepatopulmonary syndrome Hepatorenal failure Spider naevus Hepatorenal syndrome Splenorenal shunt Hepatotoxicity Intestinal varices Intestinal varices haemorrhage Varicose vein Hepatitis, non-infectious Acute graft versus host disease in liver Allergic hepatitis Chronic graft versus host disease in liver Chronic hepatitis Graft versus host disease in liver Hepatitis Hepatitis Steatohepatitis Hepatitis Hepatitis Graft versus host disease in liver Hepatitis Hepatitis Graft versus host disease in liver Hepatitis Hepatitis Graft versus host disease in liver Hepatitis cholestatic Liver sarcoidosis | Hepatocellular foamy cell syndrome | Portal shunt |
| Hepatorenal syndrome Splenorenal shunt Hepatotoxicity Splenorenal shunt procedure Intestinal varices Intestinal varices Spontaneous intrahepatic portosystemic venous shunt Intestinal varices haemorrhage Varicose vein Hepatitis, non-infectious Acute graft versus host disease in liver Allergic hepatitis Hepatitis toxic Autoimmune hepatitis Chronic graft versus host disease in liver Chronic hepatitis Chronic hepatitis Foraft versus host disease in liver Hepatitis coulce Radiation hepatitis Hepatitis Hepatitis Hepatitis Hepatitis Hepatitis Hepatitis Lupus hepatitis Graft versus host disease in liver Hepatitis Hepatitis Hepatitis Hepatitis Liver sarcoidosis | Hepatocellular injury | Portal shunt procedure |
| Hepatorenal syndrome Splenorenal shunt Hepatotoxicity Splenorenal shunt procedure Intestinal varices Spontaneous intrahepatic portosystemic venous shunt Intestinal varices haemorrhage Stomal varices Varicose vein Hepatitis, non-infectious Acute graft versus host disease in liver Allergic hepatitis Hepatitis toxic Autoimmune hepatitis Ischaemic hepatitis Chronic graft versus host disease in liver Lupus hepatitis Chronic hepatitis Schaemic hepatitis Foraft versus host disease in liver Chronic hepatitis Steatohepatitis Hepatitis Hepatitis Liver sarcoidosis Liver sarcoidosis | Hepatopulmonary syndrome | Small-for-size liver syndrome |
| Hepatotoxicity Intestinal varices Spontaneous intrahepatic portosystemic venous shunt Intestinal varices haemorrhage Varicose vein Hepatitis, non-infectious Acute graft versus host disease in liver Allergic hepatitis Autoimmune hepatitis Chronic graft versus host disease in liver Chronic hepatitis Graft versus host disease in liver Hepatitis toxic Lupus hepatitis Chronic hepatitis Non-alcoholic steatohepatitis Graft versus host disease in liver Radiation hepatitis Hepatitis Hepatitis Granulomatous liver disease Hepatitis cholestatic Liver sarcoidosis | Hepatorenal failure | Spider naevus |
| Intestinal varices Intestinal varices haemorrhage Varicose vein Hepatitis, non-infectious Acute graft versus host disease in liver Allergic hepatitis Autoimmune hepatitis Chronic graft versus host disease in liver Chronic hepatitis Graft versus host disease in liver Non-alcoholic steatohepatitis Graft versus host disease in liver Radiation hepatitis Hepatitis acute Granulomatous liver disease Liver sarcoidosis | Hepatorenal syndrome | Splenorenal shunt |
| Intestinal varices haemorrhage Varicose vein Hepatitis, non-infectious Acute graft versus host disease in liver Allergic hepatitis Autoimmune hepatitis Chronic graft versus host disease in liver Lupus hepatitis Chronic hepatitis Non-alcoholic steatohepatitis Graft versus host disease in liver Radiation hepatitis Hepatitis Hepatitis acute Granulomatous liver disease Liver sarcoidosis | Hepatotoxicity | Splenorenal shunt procedure |
| Hepatitis, non-infectious Acute graft versus host disease in liver Hepatitis fulminant Allergic hepatitis Hepatitis toxic Autoimmune hepatitis Ischaemic hepatitis Chronic graft versus host disease in liver Lupus hepatitis Chronic hepatitis Non-alcoholic steatohepatitis Graft versus host disease in liver Radiation hepatitis Hepatitis Steatohepatitis Hepatitis acute Granulomatous liver disease Hepatitis cholestatic Liver sarcoidosis | Intestinal varices | Spontaneous intrahepatic portosystemic venous shunt |
| Hepatitis, non-infectious Acute graft versus host disease in liver Hepatitis fulminant Allergic hepatitis Hepatitis toxic Autoimmune hepatitis Ischaemic hepatitis Chronic graft versus host disease in liver Lupus hepatitis Chronic hepatitis Non-alcoholic steatohepatitis Graft versus host disease in liver Radiation hepatitis Hepatitis Steatohepatitis Hepatitis acute Granulomatous liver disease Hepatitis cholestatic Liver sarcoidosis | Intestinal varices haemorrhage | Stomal varices |
| Acute graft versus host disease in liver Allergic hepatitis Autoimmune hepatitis Chronic graft versus host disease in liver Chronic hepatitis Chronic hepatitis Non-alcoholic steatohepatitis Graft versus host disease in liver Radiation hepatitis Hepatitis Steatohepatitis Hepatitis acute Granulomatous liver disease Liver sarcoidosis | Varicose vein | |
| Allergic hepatitis Autoimmune hepatitis Chronic graft versus host disease in liver Chronic hepatitis Chronic hepatitis Non-alcoholic steatohepatitis Graft versus host disease in liver Radiation hepatitis Hepatitis Steatohepatitis Hepatitis acute Granulomatous liver disease Liver sarcoidosis | Hepatitis, non-infectious | |
| Autoimmune hepatitis Chronic graft versus host disease in liver Lupus hepatitis Chronic hepatitis Non-alcoholic steatohepatitis Graft versus host disease in liver Radiation hepatitis Hepatitis Steatohepatitis Hepatitis acute Granulomatous liver disease Liver sarcoidosis | Acute graft versus host disease in liver | Hepatitis fulminant |
| Chronic graft versus host disease in liver Chronic hepatitis Chronic hepatitis Mon-alcoholic steatohepatitis Graft versus host disease in liver Radiation hepatitis Hepatitis Steatohepatitis Hepatitis acute Granulomatous liver disease Hepatitis cholestatic Liver sarcoidosis | Allergic hepatitis | Hepatitis toxic |
| Chronic hepatitis Graft versus host disease in liver Hepatitis Hepatitis acute Hepatitis cholestatic Non-alcoholic steatohepatitis Radiation hepatitis Steatohepatitis Granulomatous liver disease Liver sarcoidosis | Autoimmune hepatitis | Ischaemic hepatitis |
| Graft versus host disease in liver Hepatitis Hepatitis acute Hepatitis cholestatic Radiation hepatitis Steatohepatitis Granulomatous liver disease Liver sarcoidosis | Chronic graft versus host disease in liver | Lupus hepatitis |
| Hepatitis Steatohepatitis Hepatitis acute Granulomatous liver disease Hepatitis cholestatic Liver sarcoidosis | Chronic hepatitis | Non-alcoholic steatohepatitis |
| Hepatitis acute Granulomatous liver disease Hepatitis cholestatic Liver sarcoidosis | Graft versus host disease in liver | Radiation hepatitis |
| Hepatitis cholestatic Liver sarcoidosis | Hepatitis | Steatohepatitis |
| · | Hepatitis acute | Granulomatous liver disease |
| Hepatitis chronic active Portal tract inflammation | Hepatitis cholestatic | Liver sarcoidosis |
| | Hepatitis chronic active | Portal tract inflammation |

| 11\D\r-0000-301 | 1 uge 33 |
|---|---|
| Hepatitis chronic persistent | |
| Liver related investigations, signs and syn | nptoms |
| Alanine aminotransferase abnormal | Hypercholia |
| Alanine aminotransferase increased | Hypertransaminasaemia |
| Ammonia abnormal | Kayser-Fleischer ring |
| Ammonia increased | Liver function test abnormal |
| Ascites | Liver induration |
| Aspartate aminotransferase abnormal | Liver palpable |
| Aspartate aminotransferase increased | Liver scan abnormal |
| Bacterascites | Liver tenderness |
| Bile output abnormal | Mitochondrial aspartate aminotransferase increased |
| Bile output decreased | Molar ratio of total branched-chain amino acid to tyrosine |
| Biliary ascites | Oedema due to hepatic disease |
| Bilirubin conjugated abnormal | Perihepatic discomfort |
| Bilirubin conjugated increased | Retrograde portal vein flow |
| Bilirubin urine present | Total bile acids increased |
| Biopsy liver abnormal | Transaminases abnormal |
| Blood bilirubin abnormal | Transaminases increased |
| Blood bilirubin increased | Ultrasound liver abnormal |
| Blood bilirubin unconjugated increased | Urine bilirubin increased |
| Bromosulphthalein test abnormal | X-ray hepatobiliary abnormal |
| Child-Pugh-Turcotte score abnormal | 5'nucleotidase increased |
| Child-Pugh-Turcotte score increased | Blood alkaline phosphatase abnormal |
| Computerised tomogram liver | Blood alkaline phosphatase increased |
| Foetor hepaticus | Blood cholinesterase abnormal |
| Galactose elimination capacity test abnormal | Blood cholinesterase decreased |
| Galactose elimination capacity test decreased | Deficiency of bile secretion |
| Gamma-glutamyltransferase abnormal | Glutamate dehydrogenase increased |
| Gamma-glutamyltransferase increased | Haemorrhagic ascites |
| Guanase increased | Hepatic fibrosis marker abnormal |
| Hepaplastin abnormal | Hepatic fibrosis marker increased |
| Hepaplastin decreased | Hypoalbuminaemia |
| Hepatic artery flow decreased | Leucine aminopeptidase increased |
| Hepatic congestion | Liver function test decreased |
| Hepatic enzyme abnormal | Liver function test increased |

| Hepatic enzyme decreased | Liver iron concentration abnormal |
|---|---|
| Hepatic enzyme increased | Liver iron concentration increased |
| Hepatic function abnormal | Model for end stage liver disease score abnormal |
| Hepatic hydrothorax | Model for end stage liver disease score increased |
| Hepatic hypertrophy | Periportal oedema |
| Hepatic mass | Peritoneal fluid protein abnormal |
| Hepatic pain | Peritoneal fluid protein decreased |
| Hepatic sequestration | Peritoneal fluid protein increased |
| Hepatic vascular resistance increased | Pneumobilia |
| Hepatobiliary scan abnormal | Portal vein flow decreased |
| Hepatomegaly | Portal vein pressure increased |
| Hepatosplenomegaly | Retinol binding protein decreased |
| Hyperammonaemia | Urobilinogen urine decreased |
| Hyperbilirubinaemia | Urobilinogen urine increased |
| Hepatic disorders specifically reported as alcohol-related | |
| Alcoholic liver disease | Hepatic steato-fibrosis |
| Cirrhosis alcoholic | Hepatitis alcoholic |
| Fatty liver alcoholic | Zieve syndrome |

# CMQ LIST OF PREFERRED TERMS FOR INJECTION SITE REACTION

| Immediate post-injection reaction | Injection site ulcer |
|-----------------------------------|------------------------------------------|
| Injection related reaction | Injection site urticaria |
| Injection site abscess | Injection site vesicles |
| Injection site cellulitis | Injection site warmth |
| Injection site infection | Injection site ischaemia |
| Injection site pustule | Injection site coldness |
| Injection site abscess sterile | Injection site discolouration |
| Injection site anaesthesia | Injection site photosensitivity reaction |
| Injection site atrophy | Injection site swelling |
| Injection site bruising | Injection site discomfort |
| Injection site cyst | Injection site calcification |
| Injection site dermatitis | Injection site movement impairment |
| Injection site erosion | Injection site lymphadenopathy |
| Injection site erythema | Injection site nodule |
| Injection site extravasation | Embolia cutis medicamentosa |

| 111/1/-0000-301 | |
|---------------------------------|-------------------------------|
| Injection site fibrosis | Injection site scar |
| Injection site granuloma | Injection site discharge |
| Injection site haematoma | Injection site pallor |
| Injection site haemorrhage | Injection site papule |
| Injection site hypersensitivity | Injection site injury |
| Injection site hypertrophy | Injection site scab |
| Injection site induration | Injection site eczema |
| Injection site inflammation | Injection site streaking |
| Injection site irritation | Injection site dryness |
| Injection site mass | Injection site laceration |
| Injection site necrosis | Injection site macule |
| Injection site nerve damage | Injection site vasculitis |
| Injection site oedema | Injection site exfoliation |
| Injection site pain | Injection site dysaesthesia |
| Injection site paraesthesia | Injection site plaque |
| Injection site phlebitis | Injection site hyperaesthesia |
| Injection site pruritus | Injection site hypoaesthesia |
| Injection site rash | Injection site hypertrichosis |
| Injection site reaction | |
| Injection site thrombosis | |

# CMQ LIST OF PREFERRED TERMS FOR CNS DEPRESSION

| Mental fatigue | Hyporesponsive to stimuli |
|---|---|
| Microsleep | Benign familial neonatal convulsions |
| Narcolepsy | Febrile convulsion |
| Coma | Drug withdrawal convulsions |
| Impaired driving ability | Convulsion neonatal |
| Impaired ability to use machinery | Convulsions local |
| Accident | Tonic convulsion |
| Road traffic accident | Convulsion in childhood |
| Vision blurred | Clonic convulsion |
| Vertigo CNS origin | Acute encephalitis with refractory, repetitive partial seizures |
| Incoherent | Generalised tonic-clonic seizure |
| Disturbance in attention | Complex partial seizures |

| INDV-0000-301 | |
|---|---|
| Judgement impaired | Psychomotor seizures |
| Mental impairment | Simple partial seizures |
| Borderline mental impairment | Autonomic seizure |
| Cognitive disorder | Atonic seizures |
| Altered state of consciousness | Seizure |
| Depressed level of consciousness | Partial seizures with secondary generalisation |
| Lethargy | Alcoholic seizure |
| Loss of consciousness | Partial seizures |
| Sedation | Seizure like phenomena |
| Somnolence | Seizure cluster |
| Somnolence neonatal | Change in seizure presentation |
| Stupor | Migraine-triggered seizure |
| Syncope | Psychogenic seizure |
| Postictal state | Seizure anoxic |
| Consciousness fluctuating | Post stroke seizure |
| Neonatal oversedation | Accidental death |
| Hypoglycaemic unconsciousness | Accidental overdose |
| Hyperglycaemic unconsciousness | Accidental exposure to product |
| Post-injection delirium sedation syndrome | Cerebrovascular accident |
| Preictal state | Dizziness |
| Psychogenic pseudosyncope | Dizziness exertional |
| Mental status changes | Dizziness postural |
| Mental status changes postoperative | Procedural dizziness |
| Slow response to stimuli | Neurotoxicity |
| Unresponsive to stimuli | |

# CMQ LIST OF PREFERRED TERMS FOR RESPIRATORY DEPRESSION/RESPIRATORY FAILURE

| Acute respiratory distress syndrome | Neonatal respiratory arrest |
|-------------------------------------|----------------------------------------|
| Acute respiratory failure | Neonatal respiratory depression |
| Apnoea | Neonatal respiratory distress syndrome |
| Apnoea neonatal | Neonatal respiratory failure |
| Infantile apnoea | Respiratory arrest |
| Apnoeic attack | Respiratory depression |
| Bradypnoea | Respiratory depth decreased |

| Breath sounds absent | Respiratory distress |
|----------------------------------|------------------------------------|
| Cardio-respiratory distress | Respiratory failure |
| Central-alveolar hypoventilation | Respiratory paralysis |
| Chronic respiratory failure | Respiratory rate decreased |
| Hypopnoea | Severe acute respiratory syndrome |
| Hypoventilation | Cardio-respiratory arrest |
| Hypoventilation neonatal | Cardio-respiratory arrest neonatal |
| Lung hypoinflation | Cardiopulmonary failure |
| Meconium aspiration syndrome | |

# CMQ LIST OF PREFERRED TERMS FOR ORTHOSTATIC HYPOTENSION

| Orthostatic hypotension | Syncope |
|-------------------------|-----------------------|
| Vision blurred | Presyncope |
| Dizziness | Diastolic hypotension |
| Dizziness exertional | Hypotension |
| Dizziness postural | |

# CMQ LIST OF PREFERRED TERMS FOR WITHDRAWAL SYMPTOMS

| Agitation | Malaise |
|------------------------|----------------------------|
| Anxiety | Muscle spasms |
| Arthralgia | Muscle twitching |
| Bone pain | Myalgia |
| Chills | Mydriasis |
| Decreased appetite | Nausea |
| Depression | Piloerection |
| Diarrhoea | Pruritus |
| Dizziness | Psychomotor hyperactivity |
| Drug dependence | Pyrexia |
| Flushing | Respiratory rate increased |
| Heart rate increased | Restlessness |
| Hyperhidrosis | Rhinitis |
| Hypertension | Rhinorrhoea |
| Hypervigilance | Sneezing |
| Influenza like illness | Tachycardia |

| Insomnia | Tremor |
|-----------------------|--------------------------|
| Irritability | Vomiting |
| Lacrimal disorder | Yawning |
| Lacrimation increased | Drug withdrawal symptoms |
| Muscle strain | |

# CMQ LIST OF PREFERRED TERMS FOR ACUTE PANCREATITIS

| Amylase abnormal | Oedematous pancreatitis |
|---------------------------------------------|--------------------------------|
| Amylase creatinine clearance ratio abnormal | Pancreatic abscess |
| Amylase increased | Pancreatic enzyme abnormality |
| Bilirubin conjugated abnormal | Pancreatic enzymes abnormal |
| Blood bilirubin increased | Pancreatic enzymes increased |
| Blood trypsin increased | Pancreatic haemorrhage |
| Cullen's sign | Pancreatic necrosis |
| Grey Turner's sign | Pancreatic phlegmon |
| Haemorrhagic necrotic pancreatitis | Pancreatic pseudocyst |
| Hereditary pancreatitis | Pancreatic pseudocyst drainage |
| Hyperamylasaemia | Pancreatitis |
| Hyperbilirubinaemia | Pancreatitis acute |
| Hyperlipasaemia | Pancreatitis haemorrhagic |
| Ischaemic pancreatitis | Pancreatitis necrotising |
| Lipase abnormal | Pancreatitis relapsing |
| Lipase increased | Pancreatorenal syndrome |
| Lipase urine increased | |

## 23.2 APPENDIX 2: LIST OF CYP3A4 INHIBITOR MEDICATIONS

| Generic/Brand Name | Category | Generic/Brand Name | Category |
|--------------------|----------|--------------------|----------|
| Alprazolam | weak | isoniazid | weak |
| Amiodarone | weak | istradefylline | weak |
| Amlodipine | weak | Itraconazole | strong |
| Amprenavir | moderate | ivacaftor | weak |
| Aprepitant | moderate | Ketoconazole | strong |
| Atazanavir | moderate | lapatinib | weak |
| Atorvastatin | weak | lomitapide | weak |
| Bicalutamide | weak | lopinavir | strong |

| INDV-0000-301 | • | 1 | 1 age 39 |
|------------------------|--------------|----------------|--------------|
| boceprevir | strong | Mestranol | weak |
| Chloramphenicol | unclassified | Metronidazole | unclassified |
| chlorzoxazone | weak | Mibefradil | strong |
| cilostazol | weak | Miconazole | unclassified |
| Cimetidine | moderate | Mifepristone | unclassified |
| Ciprofloxacin | moderate | Nefazodone | strong |
| Clarithromycin | strong | Nelfinavir | strong |
| Clotrimazole | moderate | Nicardipine | unclassified |
| cobicistat | strong | nilotinib | weak |
| conivaptan | strong | Norfloxacin | unclassified |
| crizotinib | moderate | Norfluoxetine | unclassified |
| Cyclosporine | moderate | ombitasvir | strong |
| danoprevir | strong | paritaprevir | strong |
| darunavir | moderate | pazopanib | weak |
| dasabuvir | strong | posaconazole | strong |
| Delavirdine | strong | Progestogen | weak |
| Diethyldithiocarbamate | unclassified | Propofol | unclassified |
| Diltiazem | strong | Quinine | unclassified |
| dronedarone | moderate | Ranitidine | weak |
| elvitegravir | strong | ranolazine | weak |
| Erythromycin | moderate | Ritonavir | strong |
| estradiol | weak | Saquinavir | strong |
| ethinyl | weak | Sertraline | unclassified |
| Fluconazole | moderate | Starfruit | unclassified |
| Fluoxetine | weak | tacrolimus | weak |
| Fluvoxamine | moderate | Telaprevir | strong |
| fosamprenavir | moderate | Telithromycin | strong |
| fosaprepitant | weak | ticagrelor | weak |
| Gestodene | weak | tipranavir | strong |
| ginkgo | weak | tofisopam | moderate |
| goldenseal | weak | troleandomycin | strong |
| grapefruit | strong | Verapamil | moderate |
| idelalisib | strong | voriconazole | strong |

NDV-6000-301 Page 60

#### 23.3 APPENDIX 3: TABLES, FIGURES AND LISTINGS

#### Tables

#### 14.1 Demographic Data Tables & Figures

- Table 14.1.1.1 Subject Disposition All Screened Subjects
- Table 14.1.1.2 Enrollment by Site All Screened Subjects
- Table 14.1.1.3 Enrollment by Site Safety Analysis Set
- Table 14.1.1.4 Subject Analysis Sets All Screened Subjects
- Table 14.1.2.1 Demographic and Baseline Characteristics Safety Analysis Set
- Table 14.1.3.1 Medical History Safety Analysis Set
- Table 14.1.4.1 Substance Use Safety Analysis Set
- Table 14.1.5.1 Summary of Prior Medications Safety Analysis Set
- Table 14.1.5.2 Summary of Concomitant Medications during RBP-6000 Dosing Safety Analysis Set
- Table 14.1.5.3 Summary of Concomitant Medications post RBP-6000 Dosing-Safety Analysis Set
- Table 14.1.5.4 Summary of Subjects Who have taken CNS Depressant Medications during RBP-6000 Dosing (using Concomitant medication data and Urine Drug Screening) Safety Analysis Set
- Table 14.1.5.5 Summary of CNS Depressant Medications Taken during RBP-6000 dosing Safety Analysis Set
- Table 14.1.5.6 Summary of CYP3A4 Inhibitor Medications by Category (Unclassified, Weak, Moderate or Strong inhibitors) during RBP-6000 dosing Safety Analysis Set
- Table 14.1.5.7 Summary of CYP3A4 Inhibitor Medications by Category (Unclassified, Weak, Moderate or Strong inhibitors) post RBP-6000 dosing Safety Analysis Set
- Table 14.1.6.1 Summary of RBP-6000 Exposure Safety Analysis Set
- Table 14.1.6.2 Cumulative Frequency Distribution of RBP-6000 Exposure Safety Analysis Set
- Table 14.1.6.3 Summary of RBP-6000 Injections Safety Analysis Set
- Table 14.1.6.4 Cumulative Frequency Distribution of RBP-6000 Injections Safety Analysis Set
- Table 14.1.6.5 Dose Level Over Time During the Treatment Period Safety Analysis Set
- Table 14.1.6.6 Dose Level Over Time During the Treatment Period for Subjects Who Received 100 mg at the First Injection Safety Analysis Set
- Table 14.1.6.7 Dose Level Over Time During the Treatment Period for Subjects Who Received 300 mg at the First Injection Safety Analysis Set
- Table 14.1.6.8 Dose Modification and its Reason Over Time During the Treatment Period Safety Analysis Set
- Figure 14.1.6.8 Stacked Bar Chart of Dose Modification Over Time During the Treatment Period Safety Analysis Set
- Table 14.1.6.9 Frequency Distribution of Total Number of Injections in the Treatment Period by Dose Level Safety Analysis Set
- Table 14.1.6.10 Frequency Distribution of Days Since Last Injection During the Treatment Period Safety Analysis Set Figure 14.1.6.10 Distribution of Actual Injection Days Over Time During the Treatment Period Safety Analysis Set

#### 14.2 Efficacy Data Tables

- Table 14.2.1.1 Cumulative Distribution Function of the Percentage of Urine Samples Negative for Opioids in the treatment period Safety Analysis Set
- Table 14.2.1.2 Number and Percentage of Subjects with Urine Samples Negative for Opioids by Visit Safety Analysis Set
- Table 14.2.1.3 Urine Toxicology for Drug Usage for All Visits in the Treatment Period Safety Analysis Set

#### 14.3 Safety Data Tables & Figures

- Table 14.3.1.1 Overall Summary of Treatment-Emergent Adverse Events Safety Analysis Set
- Table 14.3.1.2 Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term During the Treatment Period Safety Analysis Set
- Table 14.3.1.3 Summary of Treatment-Emergent Adverse Events Experienced by >=5% of Subjects by MedDRA Preferred Term During Treatment Period—Safety Analysis Set


Table 14.3.14 Summary of Treatment-Emergent Adverse Events Leading to Discontinuation by MedDRA System Organ Class and Preferred Term During Treatment Period- Safety Analysis Set

Table 14.3.1.5 Summary of Deaths due to Adverse Event (AE) - Safety Analysis Set

Table 14.3.1.6 Summary of Serious Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term During Treatment Period—Safety Analysis Set

Table 14.3.1.7 Summary of Serious Treatment-Emergent Adverse Events Related to Study Treatment by MedDRA System Organ Class and Preferred Term During Treatment Period – Safety Analysis Set

Table 14.3.1.8 Summary of Treatment-Emergent Adverse Events by Maximum Severity, MedDRA System Organ Class and Preferred Term During Treatment Period – Safety Analysis Set

Table 14.3.1.9 Summary of Treatment-Emergent Adverse Events Related to Study Treatment by Maximum Severity, MedDRA System Organ Class and Preferred Term During the Treatment Period- Safety Analysis Set

Table 14.3.1.10 Summary of Severe Treatment-Emergent Adverse Events Related to Study Treatment Leading to Discontinuation by MedDRA System Organ Class and Preferred Term During the Treatment Period- Safety Analysis Set Table 14.3.1.11 Summary of Severe Treatment-Emergent Adverse Events by MedDRA System Organ Class and

Table 14.3.1.12 Summary of Treatment-Emergent Adverse Events Potentially Pertaining to Drug Withdrawal Symptoms by MedDRA System Organ Class and Preferred Term During the Treatment Period- Safety Analysis Set Table 14.3.1.13 Summary of Treatment-emergent Adverse Events Potentially Pertaining to Drug Withdrawal

Symptoms During the Safety Follow-up Period for Subjects Who Entered into the Safety Follow-up Period

Table 14.3.1.14 Summary of Treatment-Emergent Adverse Events Potentially Pertaining to Injection Site Reactions by MedDRA System Organ Class and Preferred Term During the Treatment Period- Safety Analysis Set

Table 14.3.1.15 Summary of Treatment-Emergent Adverse Events Potentially Pertaining to Acute Pancreatitis by MedDRA System Organ Class and Preferred Term during the Treatment Period - Safety Analysis Set

Table 14.3.1.16 Summary of Treatment-Emergent Adverse Events Potentially Pertaining to Hepatic Disorders by MedDRA System Organ Class and Preferred Term during the Treatment Period - Safety Analysis Set

Table 14.3.1.17 Summary of Treatment-Emergent Adverse Events Potentially Pertaining to Respiratory Depression and Failure by MedDRA System Organ Class and Preferred Term during the Treatment Period - Safety Analysis Set

 ${\sf Table~14.3.1.18~Summary~of~Treatment-Emergent~Adverse~Events~Potentially~Pertaining~to~Central~Nervous~System}$ 

Depression by MedDRA System Organ Class and Preferred Term during the Treatment Period - Safety Analysis Set Table 14.3.1.19 Summary of Treatment-Emergent Adverse Events Potentially Pertaining to Orthostatic Hypotension

by MedDRA System Organ Class and Preferred Term during the Treatment Period - Safety Analysis Set

Table 14.3.1.20 Summary of Treatment-Emergent Adverse Events Regarding Psychiatry History Topic by MedDRA System Organ Class and Preferred Term during the Treatment Period - Safety Analysis Set

Table 14.3.2.1 Early Removal of Study Drug Depot — Safety Analysis Set

Preferred Term During the Treatment Period- Safety Analysis Set

Table 14.3.3.1 Summary of Local Injection Site Tolerability Reactions During the Treatment Period- Safety Analysis Set Figure 14.3.3.1 Percentage of Subjects Who Reported Local Injection Site Tolerability Reactions: Pain - Safety Analysis Set

Table 14.3.3.2 Summary of Local Injection Site Visual Analog Scale (VAS) Pain Scores - Safety Analysis Set

Figure 14.3.3.2 Mean Value of Local Injection Site Visual Analog Scale (VAS) Pain Scores by visit - Safety Analysis Set

Table 14.3.3.3 Summary of Local Injection Site Burning/Stinging Evaluation - Safety Analysis Set

Table 14.3.3.4 Summary of Injection Site Evaluation During the Treatment Period: Attempted Removal - Safety Analysis Set

Table 14.3.4.1 Incidence of Columbia Suicide Severity Rating Scale (C-SSRS): Suicidal Ideation and Suicidal Behavior - Safety Analysis Set

Table 14.3.4.2 Shift Table to Demonstrate Change in C-SSRS Categories from Baseline Lifetime During the Treatment Period - Safety Analysis Set

Table 14.3.4.3 Shift Table to Demonstrate Change in C-SSRS Categories from Baseline 6 months During the Treatment Period - Safety Analysis Set

Table 14.3.4.4 Shift Table to Demonstrate Change in C-SSRS Scores from Baseline lifetime During the Treatment Period - Safety Analysis Set

Table 14.3.4.5 Shift Table to Demonstrate Change in C-SSRS Scores from Baseline 6 months During the Treatment Period - Safety Analysis Set

#### 14.3.5 Laboratory Data Tables

Table 14.3.5.1 Summary of Laboratory Data by Visit: Hematology - Safety Analysis Set

Table 14.3.5.2 Summary of Laboratory Data by Visit: Serum Chemistry - Safety Analysis Set

Table 14.3.5.3 Summary of Laboratory Data by Visit: Urinalysis - Safety Analysis Set

Table 14.3.5.4 Summary of Potential Hepatotoxicity by Visit: Serum Chemistry - Safety Analysis Set

Figure 14.3.5.4.1 Evaluation of Drug-Induced Serious Hepatotoxicity: Plot of Peak Total Bilirubin [x ULN] vs. Peak

Aspartate Aminotransferase [x ULN] on a log/log scale During the Treatment Period – Safety Analysis Set

Figure 14.3.5.4.2 Evaluation of Drug-Induced Serious Hepatotoxicity: Plot of Peak Total Bilirubin [x ULN] vs. Peak

Alanine Aminotransferase [x ULN] on a log/log scale During the Treatment Period – Safety Analysis Set

Figure 14.3.5.4.3 Evaluation of Drug-Induced Serious Hepatotoxicity: Box Plot to Assess Clinical Liver Safety Data by maximum Change from Baseline at Any Time During the Treatment Period – Safety Analysis Set

Table 14.3.5.5 Summary of Observed Laboratory Data: Shift from Baseline: Hematology - Safety Analysis Set

Table 14.3.5.6 Summary of Observed Laboratory Data: Shift from Baseline: Serum Chemistry – Safety Analysis Set

Table 14.3.5.7 Summary of Observed Laboratory Data: Shift from Baseline: Urinalysis - Safety Analysis Set

Table 14.3.5.8 Summary of Vital Signs by Visit – Observed Value and Change from Baseline – Safety Analysis Set

Table 14.3.5.9 Body Weight, BMI, Waist Circumference, Hip Circumference and Waist-to-Hip Ratio – Observed Value – Safety Analysis Set

#### Listings

Listing 16.2.1 Subject Analysis Sets, Disposition, Completion of Study/Discontinuation from Study – All Screened **Subjects** 

Listing 16.2.2 Inclusion/Exclusion Criteria

Listing 16.2.3 Inclusion/Exclusion Criteria Not Met – Screen Failure subjects

Listing 16.2.4 Important Protocol Deviations – Safety Analysis Set

Listing 16.2.5 Demographic and Baseline Characteristics – All Screened Subjects

Listing 16.2.6 Medical/Surgical History – Safety Analysis Set

Listing 16.2.7 Substance Use History – Safety Analysis Set

Listing 16.2.8 Study Drug Injection and Dosing – Safety Analysis Set

Listing 16.2.9 Dose Adjustments – Safety Analysis Set

Listing 16.2.10 Prior Medications – Safety Analysis Set

Listing 16.2.11.1 Concomitant Medications During RBP-6000 Dosing - Safety Analysis Set

Listing 16.2.11.2 Concomitant Medications Post RBP-6000 Dosing - Safety Analysis Set

Listing 16.2.12 Counseling and Behavioral Therapy – Safety Analysis Set

Listing 16.2.13 Deaths During the Study – All Screened Subjects

Listing 16.2.14 Serious Adverse Events During the Study – All Screened Subjects

Listing 16.2.15 Adverse Events During the Study – All Screened Subjects

Listing 16.2.16 Adverse Events Leading to Discontinuation During the Treatment Period – Safety Analysis Set

Listing 16.2.17 Local Injection Site Tolerability – Safety Analysis Set

Listing 16.2.18 Severe/Life Threatening Local Injection Site Tolerability Results and Corresponding Visual Analog Scale (VAS) Scores – Safety Analysis Set

Listing 16.2.19 Local Injection Site Visual Analog Scale (VAS) Pain Scores - Safety Analysis Set

Listing 16.2.20 Local Injection Site Burning/Stinging Evaluation – Safety Analysis Set

Listing 16.2.21 Injection Site Evaluation: Attempted Removal – Safety Analysis Set


Listing 16.2.22 Columbia Suicide Severity Rating Scale (C-SSRS): Suicidal Ideation and Behavior – Safety Analysis Set

Listing 16.2.23 Columbia Suicide Severity Rating Scale (C-SSRS): Suicidal Ideation Scores – Safety Analysis Set

Listing 16.2.24 Columbia Suicide Severity Rating Scale (C-SSRS): Suicidal Ideation Intensity Rating – Safety Analysis Set (Subjects with a Suicidal Ideation)

Listing 16.2.25 Treatment-Emergent Adverse Events Leading to Dose Reduction During the Treatment Period – Safety Analysis Set

Listing 16.2.26 Laboratory Data: Hematology – Safety Analysis Set

Listing 16.2.27 Laboratory Data: Serum Chemistry – Safety Analysis Set

Listing 16.2.28 Laboratory Data: Urinalysis - Safety Analysis Set

Listing 16.2.29 Screening Laboratory Data—Safety Analysis Set

Listing 16.2.30 Urine Drug Screening – Safety Analysis Set

Listing 16.2.31 Urine Pregnancy Test – Safety Analysis Set

Listing 16.2.32 Subjects Who Met Potential Hepatotoxicity Criteria – Safety Analysis Set

Listing 16.2.33 Laboratory Data for Subjects Who Met Potential Hepatotoxicity Criteria (Any Time Post Baseline)—Safety Analysis Set

Listing 16.2.34 Vital Signs – Safety Analysis Set

Listing 16.2.35 Body Weight, BMI, Waist Circumference, Hip Circumference and Waist-to-Hip Ratio – Safety Analysis Set

Listing 16.2.36 Listing of Actual Injection Days Over Time During the Treatment Period – Safety Analysis Set